CLINICAL TRIAL: NCT04762680
Title: Immunogenicity and Safety of SARS-CoV-2 Recombinant Protein Vaccines With AS03 Adjuvant in Adults 18 Years of Age and Older as a Primary Series and Immunogenicity and Safety of a Booster Dose of SARS-CoV-2 Adjuvanted Recombinant Protein Vaccines (Two Monovalent and One Bivalent)
Brief Title: Study of Recombinant Protein Vaccines With Adjuvant as a Primary Series and as a Booster Dose Against COVID-19 in Adults 18 Years of Age and Older
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAT00002; U1111-1251-4616 (Registry Identifier: ICTRP); 2020-003370-41 (EudraCT Number)
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: To address the emergence of variant strains, Sanofi Pasteur is developing monovalent and bivalent vaccines for use as universal late booster vaccines which will be studied in additional Phase 3 study cohorts that are added to the initial Phase 2 protocol cohorts. Supplemental Cohorts 1 and 2 will evaluate booster vaccine candidates.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In the original Phase 2 part, participants, outcome assessors, Investigators, laboratory personnel, and sponsor study staff are blinded to intervention group; and those preparing the study interventions are unblinded to vaccine assignment group.
  The supplemental Cohort 1 intervention group and Supplemental Cohorts Comparator Group will be open-label. Supplemental Cohort 2 will involve sequential randomization to main arms then exploratory arms, and the intervention will be modified double-blind (observer-blinded, as described).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Phase 2 Cohort -SARS-CoV-2 vaccine Formulation 1 (Experimental): 2 injections of SARS-CoV-2 vaccine Formulation 1 at Day 1 and Day 22
  Interventions: Biological: SARS-CoV-2 recombinant protein vaccine Phase 2 Formulation 1
- Phase 2 Cohort - SARS-CoV-2 vaccine Formulation 2 (Experimental): 2 injections of SARS-CoV-2 vaccine Formulation 2 at Day 1 and Day 22
  Interventions: Biological: SARS-CoV-2 recombinant protein vaccine Phase 2 Formulation 2
- Phase 2 Cohort - SARS-CoV-2 vaccine Formulation 3 (Experimental): 2 injections of SARS-CoV-2 vaccine Formulation 3 Day 1 and Day 22
  Interventions: Biological: SARS-CoV-2 recombinant protein vaccine Phase 2 Formulation 3
- Supplemental Cohort 1 - Booster Monovalent (D614)-AS03 SARS-CoV-2 vaccine (Experimental): Participants who were previously vaccinated 4 to < 10 months prior with an authorized mRNA or adenovirus-vector COVID-19 vaccine will receive 1 booster injection of monovalent (D614)-AS03 SARS-CoV-2 vaccine
  Interventions: Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine, monovalent (D614)-AS03, Dosage A
- Supplemental Cohort 2 - Booster Monovalent (B.1.351)-AS03 SARS-CoV-2 vaccine (Experimental): Participants who were vaccinated 4 to < 10 months prior with an authorized mRNA or adenovirus-vector COVID-19 vaccine or SARS-Cov-2 vaccine will receive 1 booster injection of monovalent (B.1.351)-AS03 SARS-CoV-2 vaccine
  Interventions: Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine, monovalent (B.1.351)-AS03
- Supplemental Cohort 2 - Booster Bivalent (D614 + B.1.351)-AS03 SARS-CoV-2 vaccine (Experimental): Participants who were vaccinated 4 to < 10 months prior with an authorized mRNA or adenovirus-vector COVID-19 vaccine will receive 1 booster injection of bivalent (D614+B.1.351)-AS03 SARS-CoV-2 vaccine
  Interventions: Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine, bivalent (D614+B.1.351)-AS03
- Supplemental Cohort 2 - Booster Monovalent (D614)-AS03 SARS-CoV-2 vaccine (Experimental): Participants who were vaccinated 4 to < 10 months prior with SARS-Cov-2 vaccine will receive 1 booster injection of monovalent (D614)-AS03 SARS-CoV-2 vaccine
  Interventions: Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine, monovalent (D614)-AS03, Dosage A
- Supplemental Comparator for Cohort 1 and 2 Boosters - Monovalent (D614)-AS03 SARS-CoV-2 vaccine (Active Comparator): 2 injections of monovalent (D614)-AS03 SARS-CoV-2 vaccine at Day 1 and Day 22 in previously unvaccinated, naïve participants
  Interventions: Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine, monovalent (D614)-AS03, Dosage B
- Cohort 2 - Booster Exploratory 1 (Experimental): Participants who were vaccinated 4 to < 10 months prior with an authorized mRNA COVID-19 vaccine will receive 1 booster injection of monovalent (B.1.351)-AS03 SARS-CoV-2 vaccine
  Interventions: Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine, monovalent (B.1.351)-AS03 Alternative Exploratory Formulation 1
- Cohort 2 - Booster Exploratory 2 (Experimental): Participants who were vaccinated 4 to < 10 months prior with an authorized mRNA COVID-19 vaccine will receive 1 booster injection of monovalent (B.1.351)-AS03 SARS-CoV-2 vaccine
  Interventions: Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine, monovalent (B.1.351)-AS03 Alternative Exploratory Formulation 2
- Cohort 2 - Booster Exploratory 3 (Experimental): Participants who were vaccinated 4 to < 10 months prior with an authorized mRNA COVID-19 vaccine will receive 1 booster injection of monovalent (B.1.351)-AS03 SARS-CoV-2 vaccine
  Interventions: Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine, monovalent (B.1.351)-AS03 Alternative Exploratory Formulation 3
- Cohort 2 - Booster Exploratory 4 (Experimental): Participants who were vaccinated 4 to < 10 months prior with an authorized mRNA COVID-19 vaccine will receive 1 booster injection of monovalent (B.1.351)-AS03 SARS-CoV-2 vaccine
  Interventions: Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine, monovalent (B.1.351)-AS03 Alternative Exploratory Formulation 4

INTERVENTIONS:
Biological: SARS-CoV-2 recombinant protein vaccine Phase 2 Formulation 1 — Pharmaceutical form: Emulsion for injection Route of administration: Intramuscular injection
  Other Names: rSP-COVID19
  Arms: Phase 2 Cohort -SARS-CoV-2 vaccine Formulation 1
Biological: SARS-CoV-2 recombinant protein vaccine Phase 2 Formulation 2 — Pharmaceutical form: Emulsion for injection Route of administration: Intramuscular injection
  Other Names: rSP-COVID19 Formulation 2
  Arms: Phase 2 Cohort - SARS-CoV-2 vaccine Formulation 2
Biological: SARS-CoV-2 recombinant protein vaccine Phase 2 Formulation 3 — Pharmaceutical form: Emulsion for injection Route of administration: Intramuscular injection
  Other Names: rSP-COVID19 Formulation 3
  Arms: Phase 2 Cohort - SARS-CoV-2 vaccine Formulation 3
Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine, monovalent (D614)-AS03, Dosage A — Pharmaceutical form: Emulsion for injection Route of administration: Intramuscular injection
  Other Names: rSP-COVID19 (D614)-AS03, Dosage A
  Arms: Supplemental Cohort 1 - Booster Monovalent (D614)-AS03 SARS-CoV-2 vaccine; Supplemental Cohort 2 - Booster Monovalent (D614)-AS03 SARS-CoV-2 vaccine
Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine, monovalent (B.1.351)-AS03 — Pharmaceutical form: Emulsion for injection Route of administration: Intramuscular injection
  Other Names: rSP-COVID19 (B.1.351)-AS03
  Arms: Supplemental Cohort 2 - Booster Monovalent (B.1.351)-AS03 SARS-CoV-2 vaccine
Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine, monovalent (D614)-AS03, Dosage B — Pharmaceutical form: Emulsion for injection Route of administration: Intramuscular injection
  Other Names: rSP-COVID19 (D614)-AS03, Dosage B
  Arms: Supplemental Comparator for Cohort 1 and 2 Boosters - Monovalent (D614)-AS03 SARS-CoV-2 vaccine
Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine, monovalent (B.1.351)-AS03 Alternative Exploratory Formulation 1 — Pharmaceutical form: Emulsion for injection Route of administration: Intramuscular injection
  Other Names: rSP-COVID19 (B.1.351)-AS03 Alternative Exploratory Formulation 1
  Arms: Cohort 2 - Booster Exploratory 1
Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine, monovalent (B.1.351)-AS03 Alternative Exploratory Formulation 2 — Pharmaceutical form: Emulsion for injection Route of administration: Intramuscular injection
  Other Names: rSP-COVID19 (B.1.351)-AS03 Alternative Exploratory Formulation 2
  Arms: Cohort 2 - Booster Exploratory 2
Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine, monovalent (B.1.351)-AS03 Alternative Exploratory Formulation 3 — Pharmaceutical form: Emulsion for injection Route of administration: Intramuscular injection
  Other Names: rSP-COVID19 (B.1.351)-AS03 Alternative Exploratory Formulation 3
  Arms: Cohort 2 - Booster Exploratory 3
Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine, monovalent (B.1.351)-AS03 Alternative Exploratory Formulation 4 — Pharmaceutical form: Emulsion for injection Route of administration: Intramuscular injection
  Other Names: rSP-COVID19 (B.1.351)-AS03 Alternative Exploratory Formulation 4
  Arms: Cohort 2 - Booster Exploratory 4
Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine, bivalent (D614+B.1.351)-AS03 — Pharmaceutical form: Emulsion for injection Route of administration: Intramuscular injection
  Other Names: rSP-COVID19 (D614+B.1.351)-AS03
  Arms: Supplemental Cohort 2 - Booster Bivalent (D614 + B.1.351)-AS03 SARS-CoV-2 vaccine

SUMMARY:
The primary objectives of the study are:

To assess the safety profile of the study vaccines in each study intervention group.

To assess the neutralizing antibody profile after primary series vaccination in SARS-CoV-2-naïve adults.

To demonstrate that a booster dose of monovalent or bivalent SARS-CoV-2 vaccine given to adults previously vaccinated with an authorized/approved COVID-19 vaccine induces an immune response that is non-inferior to the response induced by a twodose priming series with the monovalent vaccine, and superior to that observed immediately before booster.

The secondary objectives of the study are:

To assess the neutralizing and binding antibody profiles after primary series vaccination at pre-defined time points during the study.

To assess the neutralizing and binding antibody responses of booster vaccination.

To describe the occurrences of laboratory-confirmed symptomatic COVID19 after primary series and booster vaccination.

To describe the occurrences of serologically-confirmed SARS-CoV-2 infection after primary series vaccination.

DETAILED DESCRIPTION:
The duration of each participant's participation in the study will be approximately:

Original Phase 2 part: 365 days postinjection 2 (ie, 386 days total). Supplemental Cohorts 1 and 2: 365 days post-booster injection (ie, 366 days total).

ELIGIBILITY:
Inclusion Criteria:

-Aged 18 years or older on the day of inclusion. - -A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies: Is of non-childbearing potential. To be considered of non-childbearing potential, a female mut be post-menopausal for at least 1 year or surgically sterile.

OR Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to the first vaccination until at least 12 weeks after the last vaccination (ie, second dose of primary series or booster injection). A participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) within 4 hours before any dose of study intervention. - -Informed consent form has been signed and dated.

Able to attend all scheduled visits and to comply with all study procedures. SARS-CoV-2 rapid serodiagnostic test performed at the time of enrollment to detect presence of SARS-CoV-2 antibodies (Original Phase 2 Cohort).

For persons living with human immunodeficiency virus (HIV), stable HIV infection determined by participant currently on antiretrovirals with CD4 count > 200/mm3.

Does not intend to receive an authorized/approved COVID-19 vaccine from first vaccination to 3 weeks after the second vaccination despite encouragement by the investigator to receive the authorized vaccine available to them at the time of enrollment.

Supplemental cohorts: for participants originally enrolled in the Phase II cohort of the study, informed consent has to be signed and dated for transitioning to Supplemental Cohort 2.

Supplemental cohorts, Booster arms: received a complete primary vaccination series with an authorized/conditionally approved mRNA COVID-19 vaccine (mRNA-1273 [Moderna] or BNT162b2 [Pfizer/BioNTech]) or adenovirus-vectored COVID-19 vaccine (ChAdOx1 nCoV-19 [Oxford University/AstraZeneca] or Ad26.CoV2.S [J&J/Janssen]), with the last dose administered a minimum of 4 months prior to inclusion but not longer than 10 months prior to inclusion.

Exclusion Criteria:

-Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to a vaccine containing any of the same substances.

Dementia or any other cognitive condition at a stage that could interfere with following the trial procedures based on Investigator or designee's judgment.

Self-reported thrombocytopenia, contraindicating intramuscular (IM) vaccination based on Investigator's judgment.

Bleeding disorder, or receipt of anticoagulants in the past 21 days preceding inclusion, contraindicating IM vaccination based on Investigator's judgment.

Unstable acute or chronic illness that in the opinion of the Investigator or designee poses additional risk as a result of participation or that could interfere with the study procedures.

Receipt of solid-organ or bone marrow transplants in the past 180 days. Receipt of anti-cancer chemotherapy in the last 90 days. Receipt of immunoglobulins, blood, or blood-derived products in the past 3 months.

Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]). A prospective participant should not be included in the trial until the condition has resolved or the febrile event has subsided. Receipt of any vaccine in the 30 days preceding or on the day of the first study vaccination or planned receipt of any vaccine between the first study vaccination and in the 30 days following the second study vaccination except for influenza vaccination, which may be received at any time in relation to study intervention.

Applicable to Original Phase II Cohort, Supplemental Cohort 1 and Cohort 2 Comparator Group: Prior administration of a coronavirus vaccine (SARS-CoV-2, SARS-CoV, Middle East Respiratory Syndrome [MERS-CoV]). Participation at the time of study enrollment (or in the 30 days preceding the first study vaccination) or planned participation during the present study trial period in another clinical study investigating a vaccine, drug, medical device, or medical procedure. Exclusion criterion for the Supplemental Cohort 1 and Cohort 2 comparator group: positive rapid diagnostic test for SARS-CoV-2 antibodies at time of enrollment.

Exclusion criterion for participants in Supplemental Cohort 2 who were primed as participant in the Original Phase II Cohort of the present study: Receipt of authorized/conditionally approved COVID-19 vaccine after enrollment in Original Phase 2 Cohort.

Exclusion criterion for all Booster groups: Documented virologically-confirmed SARS-CoV-2 infection (by NAAT) after first dose of primary immunization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3159 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (66):
- United States (30):
  - Synexus - Clinical Research Advantage, Inc. Site Number : 8400270, Birmingham, Alabama
  - Synexus Chandler Site Number : 8400251, Chandler, Arizona
  - Synexus - Glendale. Site Number : 8400271, Glendale, Arizona
  - Baptist Health Center for Clinical Research Site Number : 8400077, Little Rock, Arkansas
  - Charles R. Drew University of Medicine and Science Site Number : 8400220, Los Angeles, California
  - Peninsula Research Associates, Inc. Site Number : 8400094, Rolling Hills Estates, California
  - Optimal Research Site Number : 8400173, San Diego, California
  - Yale University Site Number : 8400239, New Haven, Connecticut
  - The George Washington University Site Number : 8400212, Washington D.C., District of Columbia
  - Cenexel Research Centers of America Site Number : 8400089, Hollywood, Florida
  - Optimal Research, LLC Site Number : 8400057, Melbourne, Florida
  - Synexus Clinical Research US, Inc. - Orlando Site Number : 8400179, Orlando, Florida
  - Emory University Decatur Site Number : 8400201, Decatur, Georgia
  - Chicago Clinical Research Institute, Inc. Site Number : 8400269, Chicago, Illinois
  - Optimal Research Site Number : 8400187, Peoria, Illinois
  - Synexus Clinical Research Evansville Site Number : 8400272, Evansville, Indiana
  - Research Works INC Site Number : 8400045, New Orleans, Louisiana
  - Optimal Research, LLC Rockville Site Number : 8400048, Rockville, Maryland
  - Brigham and Women's Hospital Site Number : 8400199, Boston, Massachusetts
  - Synexus St. Louis Site Number : 8400100, St Louis, Missouri
  - Velocity Clinical Research, Omaha Site Number : 8400030, Omaha, Nebraska
  - Holy Name Medical Center Site Number : 8400072, Teaneck, New Jersey
  - NYU VC-Augustana Site Number : 8400267, Brooklyn, New York
  - New York University Langone Vaccine Center Site Number : 8400230, New York, New York
  - Columbia University Irving Medical Center Site Number : 8400203, New York, New York
  - University of Rochester Site Number : 8400207, Rochester, New York
  - University of Pittsburgh Site Number : 8400233, Pittsburgh, Pennsylvania
  - Coastal Carolina Research Center Site Number : 8400097, North Charleston, South Carolina
  - American Indian Clinical Trials Research Network Site Number : 8400204, Rapid City, South Dakota
  - AES Austin Site Number : 8400191, Austin, Texas
- Australia (5):
  - Investigational Site Number : 0360001, South Brisbane, Queensland
  - Investigational Site Number : 0360003, Norwood
  - Investigational Site Number : 0360002, Southport
  - Investigational Site Number : 0360005, Westmead
  - Investigational Site Number : 0360004, Woodville
- France (11):
  - Investigational Site Number : 2500013, Dijon
  - Investigational Site Number : 2500008, Limoges
  - Investigational Site Number : 2500014, Lyon
  - Investigational Site Number : 2500015, Marseille
  - Investigational Site Number : 2500016, Marseille
  - Investigational Site Number : 2500006, Nantes
  - Investigational Site Number : 2500005, Paris
  - Investigational Site Number : 2500003, Pessac
  - Investigational Site Number : 2500007, Pierre-Bénite
  - Investigational Site Number : 2500004, Rennes
  - Investigational Site Number : 2500002, Tours
- Honduras (2):
  - Investigational Site Number : 3400002, Municipio Del Distrito Central
  - Investigational Site Number : 3400001, San Pedro Sula
- New Zealand (5):
  - Investigational Site Number : 5540005, New Lynn, Auckland
  - Investigational Site Number : 5540002, Christchurch
  - Investigational Site Number : 5540007, Nawton
  - Investigational Site Number : 5540010, Nelson
  - Investigational Site Number : 5540001, Rotorua
- Spain (5):
  - Investigational Site Number : 7240013, Santiago de Compostela, Galicia [Galicia]
  - Investigational Site Number : 7240016, Majadahonda, Madrid
  - Investigational Site Number : 7240009, Madrid
  - Investigational Site Number : 7240008, Valencia
  - Investigational Site Number : 7240003, Vigo
- United Kingdom (8):
  - Investigational Site Number : 8260011, Runcorn, Halton
  - Investigational Site Number : 8260017, Bath, Somerset
  - Investigational Site Number : 8260013, Surrey, Sutton
  - Investigational Site Number : 8260014, Doncaster
  - Investigational Site Number : 8260016, Gloucester
  - Investigational Site Number : 8260010, Harrow
  - Investigational Site Number : 8260015, London
  - Investigational Site Number : 8260012, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] de Bruyn G, Wang J, Purvis A, Ruiz MS, Adhikarla H, Alvi S, Bonaparte MI, Brune D, Bueso A, Canter RM, Ceregido MA, Deshmukh S, Diemert D, Finn A, Forrat R, Fu B, Gallais J, Griffin P, Grillet MH, Haney O, Henderson JA, Koutsoukos M, Launay O, Torres FM, Masotti R, Michael NL, Park J, Rivera-Medina DM, Romanyak N, Rook C, Schuerman L, Sher LD, Tavares-Da-Silva F, Whittington A, Chicz RM, Gurunathan S, Savarino S, Sridhar S; VAT00002 booster cohorts study team. Safety and immunogenicity of a variant-adapted SARS-CoV-2 recombinant protein vaccine with AS03 adjuvant as a booster in adults primed with authorized vaccines: a phase 3, parallel-group study. EClinicalMedicine. 2023 Jul 22;62:102109. doi: 10.1016/j.eclinm.2023.102109. eCollection 2023 Aug. PMID 37533419
- [Derived] Sridhar S, Joaquin A, Bonaparte MI, Bueso A, Chabanon AL, Chen A, Chicz RM, Diemert D, Essink BJ, Fu B, Grunenberg NA, Janosczyk H, Keefer MC, Rivera M DM, Meng Y, Michael NL, Munsiff SS, Ogbuagu O, Raabe VN, Severance R, Rivas E, Romanyak N, Rouphael NG, Schuerman L, Sher LD, Walsh SR, White J, von Barbier D, de Bruyn G, Canter R, Grillet MH, Keshtkar-Jahromi M, Koutsoukos M, Lopez D, Masotti R, Mendoza S, Moreau C, Ceregido MA, Ramirez S, Said A, Tavares-Da-Silva F, Shi J, Tong T, Treanor J, Diazgranados CA, Savarino S. Safety and immunogenicity of an AS03-adjuvanted SARS-CoV-2 recombinant protein vaccine (CoV2 preS dTM) in healthy adults: interim findings from a phase 2, randomised, dose-finding, multicentre study. Lancet Infect Dis. 2022 May;22(5):636-648. doi: 10.1016/S1473-3099(21)00764-7. Epub 2022 Jan 25. PMID 35090638
- See also: VAT00002 Plain language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25374&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Phase 2 of study was conducted at 20 centers between 24 February 2021 and 01 May 2021. The Phase 3 of study was conducted at 110 centers between 29 July 2021 and 06 January 2023.
  CoV2 preS dTM= Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) prefusion Spike delta TM, PBP=Pfizer/BioNTech Primed, MP= Moderna Primed, OUAP= Oxford University/AstraZeneca Primed, JJJP= J&J/Janssen Primed and PP= Protein Primed.
Pre-assignment Details: 722 participants were enrolled in Phase 2 and 2647 participants (supplemental Phase 3=2617 and exploratory Phase 3=30) were enrolled in Phase 3 of the study. A total of 3159 unique participants were enrolled in the study. Participants from the Original Cohort were included in the Booster Cohorts because these assessed separate objectives. To be eligible, participants in the Booster Cohorts were required to have received a primary series, as administered in the Original Cohort.
Groups:
- Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1: Participants received CoV2 preS dTM monovalent D614 antigen dose 1 with fixed dose of AS03 adjuvant intermuscular (IM) injection once daily on Days 1 and 22.
- Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2: Participants received CoV2 preS dTM monovalent D614 antigen dose 2 with fixed dose of AS03 adjuvant IM injection once daily on Days 1 and 22.
- Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3: Participants received CoV2 preS dTM monovalent D614 antigen dose 3 with fixed dose of AS03 adjuvant IM injection once daily on Days 1 and 22.
- Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614): Participants previously vaccinated with Pfizer/BioNTech vaccine received a single booster dose of CoV2 preS dTM monovalent D614 antigen dose 1 with full-dose of AS03 adjuvant IM injection between 4 to 10 months after priming vaccine.
- Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351): Participants previously vaccinated with Pfizer/BioNTech vaccine received a single booster dose of CoV2 preS dTM monovalent B.1.351 antigen dose 1 with full-dose of AS03 adjuvant IM injection between 4 to 10 months after priming vaccine.
- Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351): Participants previously vaccinated with Pfizer/BioNTech vaccine received a single booster dose of CoV2 preS dTM monovalent D614 antigen dose 4 plus B.1.351 antigen dose 4 with full-dose of AS03 adjuvant IM injection between 4 to 10 months after priming vaccine.
- Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614): Participants previously vaccinated with Moderna vaccine received a single booster dose of CoV2 preS dTM monovalent D614 antigen dose 1 with full-dose of AS03 adjuvant IM injection between 4 to 10 months after priming vaccine.
- Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351): Participants previously vaccinated with Moderna vaccine received a single booster dose of CoV2 preS dTM monovalent B.1.351 antigen dose 1 with full-dose of AS03 adjuvant IM injection between 4 to 10 months after priming vaccine.
- Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351): Participants previously vaccinated with Moderna vaccine received a single booster dose of CoV2 preS dTM monovalent D614 antigen dose 4 plus B.1.351 antigen dose 4 with full-dose of AS03 adjuvant IM injection between 4 to 10 months after priming vaccine.
- Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614): Participants previously vaccinated with Oxford University/AstraZeneca vaccine received a single booster dose of CoV2 preS dTM monovalent D614 antigen dose 1 with full-dose of AS03 adjuvant IM injection between 4 to 10 months after priming vaccine.
- Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351): Participants previously vaccinated with Oxford University/AstraZeneca vaccine received a single booster dose of CoV2 preS dTM monovalent B.1.351 antigen dose 1 with full-dose of AS03 adjuvant IM injection between 4 to 10 months after priming vaccine.
- Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351): Participants previously vaccinated with Oxford University/AstraZeneca vaccine received a single booster dose of CoV2 preS dTM monovalent D614 antigen dose 4 plus B.1.351 antigen dose 4 with full-dose of AS03 adjuvant IM injection between 4 to 10 months after priming vaccine.
- Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614): Participants previously vaccinated with J&J/Janssen vaccine received a single booster dose of CoV2 preS dTM monovalent D614 antigen dose 1 with full-dose of AS03 adjuvant IM injection between 4 to 10 months after priming vaccine.
- Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351): Participants previously vaccinated with J&J/Janssen vaccine received a single booster dose of CoV2 preS dTM monovalent B.1.351 antigen dose 1 with full-dose of AS03 adjuvant IM injection between 4 to 10 months after priming vaccine.
- Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351): Participants previously vaccinated with J&J/Janssen vaccine received a single booster dose of CoV2 preS dTM monovalent D614 antigen dose 4 plus B.1.351 antigen dose 4 with full-dose of AS03 adjuvant IM injection between 4 to 10 months after priming vaccine.
- Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614): Participants previously vaccinated with protein based vaccine in Phase 2 of the study received a single booster dose of CoV2 preS dTM monovalent D614 antigen dose 1 with full-dose of AS03 adjuvant IM injection between 4 to 10 months after priming vaccine.
- Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351): Participants previously vaccinated with protein based vaccine in Phase 2 of the study received a single booster dose of CoV2 preS dTM monovalent B.1.351 antigen dose 1 with full-dose of AS03 adjuvant IM injection between 4 to 10 months after priming vaccine.
- Phase 3: Comparator: CoV2 preS dTM-AS03 (D614): SARS CoV 2 naïve and unvaccinated participants received CoV2 preS dTM monovalent D614 antigen dose 2 with full-dose of AS03 adjuvant IM injection once daily on Days 1 and 22.
- Phase 3: Exploratory 1: PBP - CoV2 preS dTM (B.1.351): Participants previously vaccinated with Pfizer mRNA vaccine received a single booster dose of CoV2 preS dTM monovalent B.1.351 antigen dose 4 with full-dose of AS03 adjuvant IM injection between 4 to 10 months after priming vaccine.
- Phase 3: Exploratory 2: PBP - CoV2 preS dTM (B.1.351): Participants previously vaccinated with Pfizer mRNA vaccine received a single booster dose of CoV2 preS dTM monovalent B.1.351 antigen dose 4 with half-dose of AS03 adjuvant IM injection between 4 to 10 months after priming vaccine.
- Phase 3: Exploratory 3: PBP - CoV2 preS dTM (B.1.351): Participants previously vaccinated with Pfizer mRNA vaccine received a single booster dose of CoV2 preS dTM monovalent B.1.351 antigen dose 1 with half-dose of AS03 adjuvant IM injection between 4 to 10 months after priming vaccine.
- Phase 3: Exploratory 4: PBP - CoV2 preS dTM (B.1.351): Participants previously vaccinated with Pfizer mRNA vaccine received a single booster dose of CoV2 preS dTM monovalent B.1.351 antigen dose 1 with no adjuvant IM injection between 4 to 10 months after priming vaccine.
Period: Phase 2
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3 | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614) | Phase 3: Exploratory 1: PBP - CoV2 preS dTM (B.1.351) | Phase 3: Exploratory 2: PBP - CoV2 preS dTM (B.1.351) | Phase 3: Exploratory 3: PBP - CoV2 preS dTM (B.1.351) | Phase 3: Exploratory 4: PBP - CoV2 preS dTM (B.1.351)
Started | 241 | 239 | 242 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 199 | 204 | 204 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 42 | 35 | 38 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 5 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 23 | 21 | 28 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 14 | 8 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 3
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3 | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614) | Phase 3: Exploratory 1: PBP - CoV2 preS dTM (B.1.351) | Phase 3: Exploratory 2: PBP - CoV2 preS dTM (B.1.351) | Phase 3: Exploratory 3: PBP - CoV2 preS dTM (B.1.351) | Phase 3: Exploratory 4: PBP - CoV2 preS dTM (B.1.351)
Started | 0 (Only participants started in Phase 3 are reported.) | 0 (Only participants started in Phase 3 are reported.) | 0 (Only participants started in Phase 3 are reported.) | 329 (Only participants started in Phase 3 are reported.) | 378 (Only participants started in Phase 3 are reported.) | 378 (Only participants started in Phase 3 are reported.) | 113 (Only participants started in Phase 3 are reported.) | 112 (Only participants started in Phase 3 are reported.) | 108 (Only participants started in Phase 3 are reported.) | 127 (Only participants started in Phase 3 are reported.) | 101 (Only participants started in Phase 3 are reported.) | 101 (Only participants started in Phase 3 are reported.) | 105 (Only participants started in Phase 3 are reported.) | 38 (Only participants started in Phase 3 are reported.) | 38 (Only participants started in Phase 3 are reported.) | 132 (Only participants started in Phase 3 are reported.) | 78 (Only participants started in Phase 3 are reported.) | 479 (Only participants started in Phase 3 are reported.) | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 302 | 338 | 337 | 102 | 105 | 100 | 119 | 95 | 98 | 94 | 32 | 31 | 126 | 71 | 368 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 27 | 40 | 41 | 11 | 7 | 8 | 8 | 6 | 3 | 11 | 6 | 7 | 6 | 7 | 111 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 4 | 1 | 5 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 1 | 0 | 10 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 13 | 17 | 12 | 8 | 3 | 2 | 4 | 3 | 1 | 3 | 2 | 1 | 4 | 6 | 32 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 9 | 22 | 24 | 2 | 4 | 6 | 4 | 3 | 0 | 5 | 4 | 6 | 1 | 1 | 66 | 0 | 0 | 0 | 0
Period: Phase 3 - Exploratory
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3 | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614) | Phase 3: Exploratory 1: PBP - CoV2 preS dTM (B.1.351) | Phase 3: Exploratory 2: PBP - CoV2 preS dTM (B.1.351) | Phase 3: Exploratory 3: PBP - CoV2 preS dTM (B.1.351) | Phase 3: Exploratory 4: PBP - CoV2 preS dTM (B.1.351)
Started | 0 | 0 | 0 | 0 (Only participants started in Phase 3 - Exploratory are reported.) | 0 (Only participants started in Phase 3 - Exploratory are reported.) | 0 (Only participants started in Phase 3 - Exploratory are reported.) | 0 (Only participants started in Phase 3 - Exploratory are reported.) | 0 (Only participants started in Phase 3 - Exploratory are reported.) | 0 (Only participants started in Phase 3 - Exploratory are reported.) | 0 (Only participants started in Phase 3 - Exploratory are reported.) | 0 (Only participants started in Phase 3 - Exploratory are reported.) | 0 (Only participants started in Phase 3 - Exploratory are reported.) | 0 (Only participants started in Phase 3 - Exploratory are reported.) | 0 (Only participants started in Phase 3 - Exploratory are reported.) | 0 (Only participants started in Phase 3 - Exploratory are reported.) | 0 (Only participants started in Phase 3 - Exploratory are reported.) | 0 (Only participants started in Phase 3 - Exploratory are reported.) | 0 (Only participants started in Phase 3 - Exploratory are reported.) | 4 (Only participants started in Phase 3 - Exploratory are reported.) | 8 (Only participants started in Phase 3 - Exploratory are reported.) | 9 (Only participants started in Phase 3 - Exploratory are reported.) | 9 (Only participants started in Phase 3 - Exploratory are reported.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 7 | 9 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Randomized set included all participants with a randomized group allocated by interactive response technology. Participants from the Original Cohort were included in the Booster Cohorts because these assessed separate objectives. To be eligible, participants in the Booster Cohorts were required to have received a primary series, as administered in the Original Cohort.
Groups:
- Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1: Participants received CoV2 preS dTM monovalent D614 antigen dose 1 with fixed dose of AS03 adjuvant IM injection once daily on Days 1 and 22.
- Total: Total of all reporting groups
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3 | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614) | Phase 3: Exploratory 1: PBP - CoV2 preS dTM (B.1.351) | Phase 3: Exploratory 2: PBP - CoV2 preS dTM (B.1.351) | Phase 3: Exploratory 3: PBP - CoV2 preS dTM (B.1.351) | Phase 3: Exploratory 4: PBP - CoV2 preS dTM (B.1.351) | Total
Number analyzed (Participants) | 241 | 239 | 242 | 329 | 378 | 378 | 113 | 112 | 108 | 127 | 101 | 101 | 105 | 38 | 38 | 132 | 78 | 479 | 4 | 8 | 9 | 9 | 3369
Age, Categorical [Count of Participants; unit: Participants] — Population: Participants from the Original Cohort were included in the Booster Cohorts because these assessed separate objectives. Therefore, baseline measure data reported for each Phase separately.
  Participants
    Phase 2: number analyzed (Participants) | 241 | 239 | 242 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 722
    Phase 2: <=18 years | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Phase 2: Between 18 and 65 years | 195 | 196 | 196 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 587
    Phase 2: >=65 years | 46 | 42 | 46 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 134
    Phase 3: number analyzed (Participants) | 0 | 0 | 0 | 329 | 378 | 378 | 113 | 112 | 108 | 127 | 101 | 101 | 105 | 38 | 38 | 132 | 78 | 479 | 0 | 0 | 0 | 0 | 2617
    Phase 3: <=18 years | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 9 | 0 | 0 | 0 | 0 | 17
    Phase 3: Between 18 and 65 years | 0 | 0 | 0 | 266 | 357 | 353 | 88 | 97 | 94 | 95 | 86 | 87 | 98 | 35 | 36 | 92 | 40 | 467 | 0 | 0 | 0 | 0 | 2291
    Phase 3: >=65 years | 0 | 0 | 0 | 63 | 17 | 23 | 25 | 15 | 13 | 32 | 15 | 14 | 6 | 3 | 2 | 40 | 38 | 3 | 0 | 0 | 0 | 0 | 309
    Phase 3 - Exploratory: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 8 | 9 | 9 | 30
    Phase 3 - Exploratory: <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 3 - Exploratory: Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 7 | 9 | 8 | 28
    Phase 3 - Exploratory: >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants from the Original Cohort were included in the Booster Cohorts because these assessed separate objectives. Therefore, baseline measure data reported for each Phase separately.
  Participants
    Phase 2: number analyzed (Participants) | 241 | 239 | 242 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 722
    Phase 2: Female | 123 | 114 | 122 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 359
    Phase 2: Male | 118 | 125 | 120 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 363
    Phase 3: number analyzed (Participants) | 0 | 0 | 0 | 329 | 378 | 378 | 113 | 112 | 108 | 127 | 101 | 101 | 105 | 38 | 38 | 132 | 78 | 479 | 0 | 0 | 0 | 0 | 2617
    Phase 3: Female | 0 | 0 | 0 | 181 | 208 | 199 | 68 | 60 | 64 | 59 | 42 | 48 | 63 | 19 | 20 | 64 | 38 | 215 | 0 | 0 | 0 | 0 | 1348
    Phase 3: Male | 0 | 0 | 0 | 148 | 170 | 179 | 45 | 52 | 44 | 68 | 59 | 53 | 42 | 19 | 18 | 68 | 40 | 264 | 0 | 0 | 0 | 0 | 1269
    Phase 3 - Exploratory: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 8 | 9 | 9 | 30
    Phase 3 - Exploratory: Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 8 | 6 | 20
    Phase 3 - Exploratory: Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 1 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Participants from the Original Cohort were included in the Booster Cohorts because these assessed separate objectives. Therefore, baseline measure data reported for each Phase separately.
  Participants
    Phase 2: American Indian or Alaska Native | 22 | 24 | 20 | 5 | 5 | 6 | 2 | 6 | 2 | 0 | 0 | 0 | 1 | 4 | 2 | 20 | 14 | 15 | 0 | 0 | 0 | 0 | 148
    Phase 2: Asian | 13 | 10 | 10 | 19 | 12 | 13 | 7 | 1 | 3 | 11 | 4 | 7 | 0 | 2 | 2 | 2 | 2 | 18 | 0 | 0 | 0 | 0 | 136
    Phase 2: Black or African American | 14 | 23 | 20 | 15 | 54 | 61 | 3 | 16 | 32 | 2 | 3 | 2 | 5 | 16 | 10 | 7 | 2 | 52 | 0 | 0 | 0 | 0 | 337
    Phase 2: Multiple | 5 | 2 | 4 | 1 | 6 | 6 | 1 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 8 | 0 | 0 | 0 | 0 | 39
    Phase 2: Native Hawaiian or Other Pacific Islander | 2 | 1 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 10
    Phase 2: White | 156 | 149 | 156 | 252 | 247 | 240 | 100 | 79 | 61 | 104 | 92 | 87 | 99 | 15 | 21 | 80 | 37 | 372 | 0 | 0 | 0 | 0 | 2347
    Phase 2: Missing | 29 | 30 | 30 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 89
    Phase 2: Not Reported | 0 | 0 | 0 | 33 | 44 | 49 | 0 | 1 | 6 | 10 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 3 | 4 | 7 | 8 | 9 | 179
    Phase 2: Unknown | 0 | 0 | 0 | 4 | 8 | 2 | 0 | 6 | 3 | 0 | 1 | 2 | 0 | 0 | 1 | 23 | 22 | 10 | 0 | 1 | 1 | 0 | 84
    Phase 3: number analyzed (Participants) | 0 | 0 | 0 | 329 | 378 | 378 | 113 | 112 | 108 | 127 | 101 | 101 | 105 | 38 | 38 | 132 | 78 | 479 | 0 | 0 | 0 | 0 | 2617
    Phase 3: American Indian or Alaska Native | 0 | 0 | 0 | 5 | 5 | 6 | 2 | 6 | 2 | 0 | 0 | 0 | 1 | 4 | 2 | 20 | 14 | 15 | 0 | 0 | 0 | 0 | 82
    Phase 3: Asian | 0 | 0 | 0 | 19 | 12 | 13 | 7 | 1 | 3 | 11 | 4 | 7 | 0 | 2 | 2 | 2 | 2 | 18 | 0 | 0 | 0 | 0 | 103
    Phase 3: Black or African American | 0 | 0 | 0 | 15 | 54 | 61 | 3 | 16 | 32 | 2 | 3 | 2 | 5 | 16 | 10 | 7 | 2 | 52 | 0 | 0 | 0 | 0 | 280
    Phase 3: Multiple | 0 | 0 | 0 | 1 | 6 | 6 | 1 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 8 | 0 | 0 | 0 | 0 | 28
    Phase 3: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 5
    Phase 3: White | 0 | 0 | 0 | 252 | 247 | 240 | 100 | 79 | 61 | 104 | 92 | 87 | 99 | 15 | 21 | 80 | 37 | 372 | 0 | 0 | 0 | 0 | 1886
    Phase 3: Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 3: Not Reported | 0 | 0 | 0 | 33 | 44 | 49 | 0 | 1 | 6 | 10 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 151
    Phase 3: Unknown | 0 | 0 | 0 | 4 | 8 | 2 | 0 | 6 | 3 | 0 | 1 | 2 | 0 | 0 | 1 | 23 | 22 | 10 | 0 | 0 | 0 | 0 | 82
    Phase 3 - Exploratory: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 8 | 9 | 9 | 30
    Phase 3 - Exploratory: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 3 - Exploratory: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 3 - Exploratory: Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 3 - Exploratory: Multiple | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 3 - Exploratory: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 3 - Exploratory: White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 3 - Exploratory: Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 3 - Exploratory: Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 7 | 8 | 9 | 28
    Phase 3 - Exploratory: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Secondary Outcome: Phase 2: Geometric Mean Titers of Neutralizing Antibodies Against SARS-CoV-2 D614G Strain at Days 22, 78, 134, 202, 292, and 387
Description: Neutralizing antibodies activity against SARS-CoV-2 D614G strain was measured with the neutralization assay (monogram assay) and the results were expressed as geometric mean titers.
Time Frame: Post-vaccination on Days 22, 78, 134, 202, 292, and 387
Population: The PPAS Naïve-D01+D22 is a subset of the FAS. Only participants analyzed at specific timepoint are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3
Number analyzed (Participants) | 159 | 160 | 160
titers
  Day 22 | 36.0 [29.4 to 44.2] | 39.6 [32.3 to 48.6] | 47.3 [37.8 to 59.1]
  Day 78: number analyzed (Participants) | 118 | 124 | 121
  Day 78 | 467 [361 to 606] | 558 [438 to 711] | 569 [458 to 707]
  Day 134: number analyzed (Participants) | 99 | 103 | 94
  Day 134 | 225 [160 to 318] | 249 [182 to 340] | 260 [190 to 358]
  Day 202: number analyzed (Participants) | 73 | 76 | 77
  Day 202 | 254 [158 to 408] | 344 [208 to 570] | 259 [159 to 421]
  Day 292: number analyzed (Participants) | 11 | 11 | 13
  Day 292 | 12145 [3643 to 40491] | 2518 [335 to 18928] | 804 [108 to 6014]
  Day 387: number analyzed (Participants) | 11 | 9 | 12
  Day 387 | 17837 [9491 to 33522] | 46305 [24179 to 88677] | 8353 [1414 to 49336]

2. Secondary Outcome: Phase 2: Number of Participants With >=2-Fold and >=4-Fold Rise in Serum Neutralization Antibody Titers Against SARS-CoV-2 D614G Strain at Days 22, 78, 134, 202, 292, and 387
Description: Neutralizing antibodies activity against SARS-CoV-2 D614G strain was measured with serum neutralization assay (monogram assay). Participants with neutralization antibody titers >=2-fold and >=4-fold increase from baseline (pre-vaccination) were analyzed.
Time Frame: Pre-vaccination on Day 1 and Post-vaccination on Days 22, 78, 134, 202, 292, and 387
Population: The PPAS Naïve-D01+D22 is a subset of the FAS. Only participants analyzed at specific timepoint are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3
Number analyzed (Participants) | 159 | 160 | 159
Participants
  Day 22: >=2-fold rise | 35 | 44 | 53
  Day 22: >=4-fold rise | 28 | 36 | 44
  Day 78: >=2-fold rise: number analyzed (Participants) | 116 | 123 | 117
  Day 78: >=2-fold rise | 108 | 116 | 113
  Day 78: >=4-fold rise: number analyzed (Participants) | 116 | 123 | 117
  Day 78: >=4-fold rise | 105 | 115 | 110
  Day 134: >=2-fold rise: number analyzed (Participants) | 98 | 102 | 93
  Day 134: >=2-fold rise | 85 | 87 | 82
  Day 134: >=4-fold rise: number analyzed (Participants) | 98 | 102 | 93
  Day 134: >=4-fold rise | 75 | 83 | 76
  Day 202: >=2-fold rise: number analyzed (Participants) | 72 | 75 | 77
  Day 202: >=2-fold rise | 57 | 62 | 62
  Day 202: >=4-fold rise: number analyzed (Participants) | 72 | 75 | 77
  Day 202: >=4-fold rise | 53 | 57 | 60
  Day 292: >=2-fold rise: number analyzed (Participants) | 10 | 11 | 13
  Day 292: >=2-fold rise | 10 | 10 | 11
  Day 292: >=4-fold rise: number analyzed (Participants) | 10 | 11 | 13
  Day 292: >=4-fold rise | 10 | 9 | 8
  Day 387: >=2-fold rise: number analyzed (Participants) | 10 | 9 | 12
  Day 387: >=2-fold rise | 10 | 9 | 11
  Day 387: >=4-fold rise: number analyzed (Participants) | 10 | 9 | 12
  Day 387: >=4-fold rise | 10 | 9 | 11

3. Secondary Outcome: Phase 2: Number of Responders as Determined by Neutralizing Antibody Titers Against SARS-CoV-2 D614G Strain at Days 22, 78, 134, 202, 292, and 387
Description: Responders were participants who had baseline values below LLOQ with detectable neutralization titer above assay LLOQ at each pre-defined post-vaccination time point and participants with baseline values above LLOQ with a 4-fold increase in neutralizing antibody titers at each pre-defined post-vaccination time point. Neutralizing antibodies activity against SARS-CoV-2 D614G strain was measured with serum neutralization assay (monogram assay).
Time Frame: Post-vaccination on Days 22, 78, 134, 202, 292, and 387
Population: The PPAS Naïve-D01+D22 is a subset of the FAS. Only participants analyzed at specific timepoint are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3
Number analyzed (Participants) | 159 | 160 | 159
Participants
  Day 22 | 35 | 44 | 53
  Day 78: number analyzed (Participants) | 116 | 123 | 117
  Day 78 | 108 | 116 | 113
  Day 134: number analyzed (Participants) | 98 | 102 | 93
  Day 134 | 85 | 87 | 82
  Day 202: number analyzed (Participants) | 72 | 75 | 77
  Day 202 | 57 | 62 | 62
  Day 292: number analyzed (Participants) | 10 | 11 | 13
  Day 292 | 10 | 10 | 11
  Day 387: number analyzed (Participants) | 10 | 9 | 12
  Day 387 | 10 | 9 | 11

4. Secondary Outcome: Phase 2: Geometric Mean Concentration (GMC) of Binding Antibodies Against SARS-CoV-2 D614G Strain at Days 1, 22, 36, 78, 134, 202, 292, and 387
Description: Binding antibodies activity against SARS-CoV-2 D614G strain was measured with Nexelis GCN4 S-enzyme-linked immunosorbent assay (ELISA) and the results were expressed as geometric mean titers.
Time Frame: Pre-vaccination on Day 1 and post-vaccination on Days 22, 36, 78, 134, 202, 292, and 387
Population: The PPAS Naïve-D01+D22 is a subset of the FAS. Only participants analyzed at specific timepoint are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3
Number analyzed (Participants) | 169 | 172 | 176
titers
  Day 1: number analyzed (Participants) | 166 | 170 | 175
  Day 1 | 10.3 [9.54 to 11.1] | 9.99 [9.52 to 10.5] | 10.2 [9.77 to 10.7]
  Day 22 | 103 [80.6 to 131] | 149 [119 to 187] | 228 [182 to 285]
  Day 36: number analyzed (Participants) | 165 | 167 | 171
  Day 36 | 15533 [13000 to 18560] | 17176 [14468 to 20390] | 18003 [15039 to 21550]
  Day 78: number analyzed (Participants) | 126 | 127 | 127
  Day 78 | 6572 [5469 to 7897] | 7526 [6112 to 9267] | 7133 [5848 to 8700]
  Day 134: number analyzed (Participants) | 105 | 111 | 100
  Day 134 | 2750 [2104 to 3594] | 2977 [2305 to 3846] | 2696 [2064 to 3521]
  Day 202: number analyzed (Participants) | 87 | 93 | 87
  Day 202 | 1414 [983 to 2033] | 1961 [1369 to 2809] | 1438 [978 to 2113]
  Day 292: number analyzed (Participants) | 12 | 12 | 14
  Day 292 | 40589 [10633 to 155000] | 9247 [1625 to 52615] | 5557 [1183 to 26116]
  Day 387: number analyzed (Participants) | 11 | 10 | 13
  Day 387 | 61087 [40242 to 92728] | 58674 [12370 to 278000] | 16234 [3146 to 83760]

5. Secondary Outcome: Phase 2: Number of Participants With >=2-Fold and >=4-Fold Rise in Binding Antibody Concentration Against SARS-CoV-2 D614G Strain at Days 22, 36, 78, 134, 202, 292, and 387
Description: Binding antibodies concentration against SARS-CoV-2 D614G strain was measured with Nexelis GCN4 S-ELISA assay. Participants with binding antibodies concentration >=2-fold and >=4-fold increase from baseline (pre-vaccination) were analyzed.
Time Frame: Pre-vaccination on Day 1 and Post-vaccination on Days 22, 36, 78, 134, 202, 292, and 387
Population: The PPAS Naïve-D01+D22 is a subset of the FAS. Only participants analyzed at specific timepoint are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3
Number analyzed (Participants) | 166 | 170 | 175
Participants
  Day 22: >=2-fold rise | 141 | 155 | 161
  Day 22: >=4-fold rise | 117 | 136 | 156
  Day 36: >=2-fold rise: number analyzed (Participants) | 159 | 161 | 166
  Day 36: >=2-fold rise | 159 | 160 | 165
  Day 36: >=4-fold rise: number analyzed (Participants) | 159 | 161 | 166
  Day 36: >=4-fold rise | 158 | 160 | 165
  Day 78: >=2-fold rise: number analyzed (Participants) | 121 | 125 | 124
  Day 78: >=2-fold rise | 121 | 124 | 124
  Day 78: >=4-fold rise: number analyzed (Participants) | 121 | 125 | 124
  Day 78: >=4-fold rise | 121 | 124 | 124
  Day 134: >=2-fold rise: number analyzed (Participants) | 101 | 110 | 100
  Day 134: >=2-fold rise | 101 | 109 | 100
  Day 134: >=4-fold rise: number analyzed (Participants) | 101 | 110 | 100
  Day 134: >=4-fold rise | 101 | 109 | 100
  Day 202: >=2-fold rise: number analyzed (Participants) | 85 | 92 | 87
  Day 202: >=2-fold rise | 85 | 91 | 86
  Day 202: >=4-fold rise: number analyzed (Participants) | 85 | 92 | 87
  Day 202: >=4-fold rise | 85 | 91 | 85
  Day 292: >=2-fold rise: number analyzed (Participants) | 11 | 12 | 14
  Day 292: >=2-fold rise | 11 | 12 | 14
  Day 292: >=4-fold rise: number analyzed (Participants) | 11 | 12 | 14
  Day 292: >=4-fold rise | 11 | 12 | 14
  Day 387: >=2-fold rise: number analyzed (Participants) | 10 | 10 | 13
  Day 387: >=2-fold rise | 10 | 10 | 13
  Day 387: >=4-fold rise: number analyzed (Participants) | 10 | 10 | 13
  Day 387: >=4-fold rise | 10 | 10 | 13

6. Secondary Outcome: Phase 2: Number of Responders as Determined by Binding Antibody Concentration Against SARS-CoV-2 D614G Strain at Days 22, 36, 78, 134, 202, 292, and 387
Description: Responders were participants who had baseline values below LLOQ with detectable antibody concentration above assay LLOQ at each pre-defined post-vaccination time point and participants with baseline values above LLOQ with a 4-fold increase in neutralizing antibody titers at each pre-defined post-vaccination time point. Binding antibodies concentration against SARS-CoV-2 D614G strain was measured with Nexelis GCN4 S-ELISA assay.
Time Frame: Post-vaccination on Days 22, 36, 78, 134, 202, 292, and 387
Population: The PPAS Naïve-D01+D22 is a subset of the FAS. Only participants analyzed at specific timepoint are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3
Number analyzed (Participants) | 166 | 170 | 175
Participants
  Day 22 | 139 | 154 | 161
  Day 36: number analyzed (Participants) | 159 | 161 | 166
  Day 36 | 159 | 160 | 165
  Day 78: number analyzed (Participants) | 121 | 125 | 124
  Day 78 | 121 | 124 | 124
  Day 134: number analyzed (Participants) | 101 | 110 | 100
  Day 134 | 101 | 109 | 100
  Day 202: number analyzed (Participants) | 85 | 92 | 87
  Day 202 | 85 | 91 | 86
  Day 292: number analyzed (Participants) | 11 | 12 | 14
  Day 292 | 11 | 12 | 14
  Day 387: number analyzed (Participants) | 10 | 10 | 13
  Day 387 | 10 | 10 | 13

7. Secondary Outcome: Phase 3: Cohort 1: Geometric Mean Titers of Neutralizing Antibodies Against SARS-CoV-2 D614G Strain and B.1.351 Variant at Days 29, 91, 181, and 366
Description: Neutralizing antibodies activity against SARS-CoV-2 D614G strain and B.1.351 variant was measured with the neutralization assay (monogram assay) and the results were expressed as geometric mean titers.
Time Frame: Post-vaccination on Days 29, 91, 181, and 366
Population: The PPAS is a subset of the FAS. Only participants analyzed for each parameter at specific timepoint are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614)
Number analyzed (Participants) | 311 | 106 | 117 | 96
titers
  Day 29: D614G | 5795 [5222 to 6432] | 5743 [4668 to 7065] | 4869 [4113 to 5764] | 4400 [3566 to 5430]
  Day 29: B.1.351: number analyzed (Participants) | 307 | 104 | 117 | 96
  Day 29: B.1.351 | 2078 [1844 to 2342] | 1726 [1355 to 2198] | 1790 [1452 to 2207] | 1390 [1095 to 1764]
  Day 91: D614G: number analyzed (Participants) | 249 | 91 | 86 | 84
  Day 91: D614G | 4623 [4037 to 5295] | 4879 [3774 to 6308] | 2704 [2065 to 3541] | 2509 [1954 to 3223]
  Day 91: B.1.351: number analyzed (Participants) | 248 | 90 | 83 | 83
  Day 91: B.1.351 | 1522 [1304 to 1776] | 1254 [920 to 1711] | 949 [702 to 1281] | 711 [540 to 936]
  Day 181: D614G: number analyzed (Participants) | 197 | 59 | 74 | 66
  Day 181: D614G | 7502 [6161 to 9135] | 10068 [6940 to 14605] | 2658 [1834 to 3852] | 5649 [3695 to 8635]
  Day 181: B.1.351: number analyzed (Participants) | 196 | 56 | 70 | 64
  Day 181: B.1.351 | 2328 [1827 to 2966] | 3217 [2073 to 4992] | 1035 [650 to 1648] | 1853 [1095 to 3134]
  Day 366: D614G: number analyzed (Participants) | 161 | 47 | 46 | 42
  Day 366: D614G | 10224 [8101 to 12903] | 10567 [6608 to 16898] | 2940 [1779 to 4858] | 6314 [3847 to 10361]
  Day 366: B.1.351: number analyzed (Participants) | 162 | 47 | 46 | 41
  Day 366: B.1.351 | 3419 [2572 to 4545] | 3349 [1929 to 5812] | 942 [533 to 1664] | 2233 [1267 to 3937]

8. Secondary Outcome: Phase 3: Cohort 1: Number of Participants With >=2-Fold and >=4-Fold Rise in Serum Neutralization Antibody Titers Against SARS-CoV-2 D614G Strain and B.1.351 Variant at Days 15, 29, 91, 181, and 366
Description: Neutralizing antibodies activity against SARS-CoV-2 D614G strain and B.1.351 variant was measured with serum neutralization assay (monogram assay). Participants with neutralization antibody titers >=2-fold and >=4-fold increase from baseline (pre-vaccination) were analyzed.
Time Frame: Pre-vaccination on Day 1 and Post-vaccination on Days 15, 29, 91, 181, and 366
Population: The PPAS is a subset of the FAS. Only participants analyzed for each parameter at specific timepoint are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614)
Number analyzed (Participants) | 290 | 104 | 114 | 87
Participants
  D614G; Day 15: >=2-fold rise: number analyzed (Participants) | 278 | 98 | 101 | 75
  D614G; Day 15: >=2-fold rise | 263 | 86 | 95 | 70
  D614G; Day 15: >=4-fold rise: number analyzed (Participants) | 278 | 98 | 101 | 75
  D614G; Day 15: >=4-fold rise | 252 | 70 | 87 | 66
  D614G; Day 29: >=2-fold rise: number analyzed (Participants) | 290 | 104 | 102 | 80
  D614G; Day 29: >=2-fold rise | 266 | 91 | 97 | 73
  D614G; Day 29: >=4-fold rise: number analyzed (Participants) | 290 | 104 | 102 | 80
  D614G; Day 29: >=4-fold rise | 250 | 79 | 87 | 68
  D614G; Day 91: >=2-fold rise: number analyzed (Participants) | 233 | 89 | 74 | 72
  D614G; Day 91: >=2-fold rise | 208 | 74 | 67 | 62
  D614G; Day 91: >=4-fold rise: number analyzed (Participants) | 233 | 89 | 74 | 72
  D614G; Day 91: >=4-fold rise | 187 | 57 | 58 | 56
  D614G; Day 181: >=2-fold rise: number analyzed (Participants) | 182 | 58 | 63 | 55
  D614G; Day 181: >=2-fold rise | 167 | 50 | 54 | 51
  D614G; Day 181: >=4-fold rise: number analyzed (Participants) | 182 | 58 | 63 | 55
  D614G; Day 181: >=4-fold rise | 149 | 44 | 42 | 41
  D614G; Day 366: >=2-fold rise: number analyzed (Participants) | 152 | 45 | 37 | 37
  D614G; Day 366: >=2-fold rise | 141 | 38 | 33 | 31
  D614G; Day 366: >=4-fold rise: number analyzed (Participants) | 152 | 45 | 37 | 37
  D614G; Day 366: >=4-fold rise | 129 | 34 | 28 | 31
  B.1.351; Day 15: >=2-fold rise: number analyzed (Participants) | 266 | 79 | 114 | 81
  B.1.351; Day 15: >=2-fold rise | 258 | 76 | 109 | 78
  B.1.351; Day 15: >=4-fold rise: number analyzed (Participants) | 266 | 79 | 114 | 81
  B.1.351; Day 15: >=4-fold rise | 246 | 67 | 103 | 76
  B.1.351; Day 29: >=2-fold rise: number analyzed (Participants) | 273 | 85 | 113 | 87
  B.1.351; Day 29: >=2-fold rise | 261 | 79 | 109 | 83
  B.1.351; Day 29: >=4-fold rise: number analyzed (Participants) | 273 | 85 | 113 | 87
  B.1.351; Day 29: >=4-fold rise | 245 | 70 | 103 | 80
  B.1.351; Day 91: >=2-fold rise: number analyzed (Participants) | 224 | 74 | 79 | 75
  B.1.351; Day 91: >=2-fold rise | 203 | 64 | 75 | 68
  B.1.351; Day 91: >=4-fold rise: number analyzed (Participants) | 224 | 74 | 79 | 75
  B.1.351; Day 91: >=4-fold rise | 189 | 54 | 67 | 66
  B.1.351; Day 181: >=2-fold rise: number analyzed (Participants) | 173 | 44 | 68 | 58
  B.1.351; Day 181: >=2-fold rise | 162 | 38 | 59 | 54
  B.1.351; Day 181: >=4-fold rise: number analyzed (Participants) | 173 | 44 | 68 | 58
  B.1.351; Day 181: >=4-fold rise | 145 | 38 | 51 | 46
  B.1.351; Day 366: >=2-fold rise: number analyzed (Participants) | 147 | 35 | 43 | 36
  B.1.351; Day 366: >=2-fold rise | 137 | 32 | 36 | 34
  B.1.351; Day 366: >=4-fold rise: number analyzed (Participants) | 147 | 35 | 43 | 36
  B.1.351; Day 366: >=4-fold rise | 127 | 30 | 34 | 30

9. Secondary Outcome: Phase 3: Cohorts 1, 2 and Comparator: Percentage of Participants With Seroresponse Against SARS-CoV-2 D614G Strain and B.1.351 Variant at 14 Days Post-Vaccination
Description: Seroresponse was defined as a >=4-fold rise in serum neutralization titer against SARS-CoV-2 D614G strain and B.1.351 variant (post/pre) at Day 15 or Day 36 relative to Day 0 or Day 22. Neutralizing antibodies activity against SARS-CoV-2 D614G strain and B.1.351 variant was measured with serum neutralization assay (monogram assay). Percentages are rounded off to the tenth decimal place.
Time Frame: Cohorts 1 and 2: 14 days post-vaccination on Day 1 (Day 15); Comparator: 14 days post-vaccination on Day 22 (Day 36)
Population: The PPAS is a subset of the FAS. Only participants analyzed for each parameter at specific timepoint are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614)
Number analyzed (Participants) | 278 | 315 | 320 | 98 | 92 | 91 | 114 | 87 | 91 | 81 | 31 | 33 | 99 | 64 | 301
percentage of participants
  D614G: number analyzed (Participants) | 278 | 315 | 320 | 98 | 92 | 91 | 101 | 87 | 88 | 75 | 31 | 33 | 99 | 64 | 301
  D614G | 90.6 [86.6 to 93.8] | 73.7 [68.4 to 78.4] | 75.6 [70.5 to 80.2] | 71.4 [61.4 to 80.1] | 72.8 [62.6 to 81.6] | 63.7 [53.0 to 73.6] | 86.1 [77.8 to 92.2] | 89.7 [81.3 to 95.2] | 89.8 [81.5 to 95.2] | 88.0 [78.4 to 94.4] | 58.1 [39.1 to 75.5] | 78.8 [61.1 to 91.0] | 84.8 [76.2 to 91.3] | 90.6 [80.7 to 96.5] | 99.0 [97.1 to 99.8]
  B.1.351: number analyzed (Participants) | 266 | 299 | 298 | 79 | 84 | 85 | 114 | 87 | 91 | 81 | 29 | 31 | 99 | 64 | 290
  B.1.351 | 92.5 [88.6 to 95.3] | 83.3 [78.6 to 87.3] | 82.9 [78.1 to 87.0] | 84.8 [75.0 to 91.9] | 83.3 [73.6 to 90.6] | 80.0 [69.9 to 87.9] | 90.4 [83.4 to 95.1] | 95.4 [88.6 to 98.7] | 96.7 [90.7 to 99.3] | 93.8 [86.2 to 98.0] | 75.9 [56.5 to 89.7] | 77.4 [58.9 to 90.4] | 85.9 [77.4 to 92.0] | 90.6 [80.7 to 96.5] | 86.6 [82.1 to 90.3]

10. Secondary Outcome: Phase 3: Cohorts 1 and 2: Geometric Mean Concentration of Binding Antibodies Against SARS-CoV-2 D614G Strain at Days 1, 15, 29, 91, 181, and 366
Description: Binding antibodies activity against SARS-CoV-2 D614G strain was measured with Nexelis GCN4 S-ELISA and the results were expressed as geometric mean titers.
Time Frame: Pre-vaccination on Day 1 and post-vaccination on Days 15, 29, 91, 181, and 366
Population: The PPAS is a subset of the FAS. Only participants analyzed at specific timepoint are reported. Results data was not collected for 'Phase 3-Exploratory reporting groups' because study vaccine used in exploratory arms were different from booster cohort. No participants were analyzed and thus data was not collected at Day 366 for "Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614)" reporting group.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351)
Number analyzed (Participants) | 326 | 362 | 361 | 110 | 108 | 107 | 125 | 97 | 99 | 99 | 37 | 37 | 130 | 77
titers
  Day 1 | 1888 [1687 to 2114] | 3032 [2621 to 3507] | 2580 [2228 to 2987] | 3236 [2729 to 3839] | 3285 [2534 to 4259] | 3505 [2747 to 4471] | 993 [781 to 1262] | 564 [427 to 747] | 537 [420 to 687] | 608 [457 to 809] | 2290 [1068 to 4908] | 996 [491 to 2021] | 1357 [1004 to 1834] | 969 [688 to 1365]
  Day 15: number analyzed (Participants) | 302 | 323 | 335 | 102 | 93 | 98 | 119 | 94 | 93 | 92 | 31 | 34 | 120 | 72
  Day 15 | 26710 [24337 to 29314] | 36428 [33227 to 39938] | 30892 [27925 to 34174] | 27390 [23220 to 32309] | 43611 [35852 to 53049] | 34704 [29398 to 40968] | 21654 [18927 to 24775] | 23775 [19137 to 29537] | 28783 [24417 to 33930] | 21758 [18254 to 25935] | 31067 [24221 to 39849] | 34534 [26146 to 45614] | 65824 [57576 to 75254] | 77057 [61772 to 96125]
  Day 29: number analyzed (Participants) | 312 | 334 | 341 | 107 | 98 | 101 | 118 | 94 | 92 | 97 | 34 | 31 | 124 | 71
  Day 29 | 20212 [18487 to 22097] | 33416 [30407 to 36723] | 27083 [24480 to 29964] | 23079 [19417 to 27431] | 48428 [39336 to 59623] | 41018 [34290 to 49065] | 13305 [11657 to 15186] | 16401 [13253 to 20296] | 17729 [14944 to 21034] | 14014 [11798 to 16647] | 29315 [22236 to 38647] | 24388 [17369 to 34243] | 60707 [52764 to 69845] | 65974 [53800 to 80902]
  Day 91: number analyzed (Participants) | 251 | 267 | 280 | 92 | 84 | 91 | 87 | 61 | 60 | 87 | 29 | 26 | 114 | 69
  Day 91 | 18845 [16780 to 21165] | 29384 [25972 to 33244] | 23908 [20860 to 27402] | 20758 [16506 to 26107] | 37791 [29062 to 49140] | 35363 [28656 to 43639] | 9792 [8093 to 11849] | 10365 [8105 to 13255] | 13189 [10078 to 17261] | 9032 [7387 to 11043] | 18463 [13497 to 25255] | 16236 [9684 to 27219] | 41282 [34967 to 48736] | 40566 [32032 to 51373]
  Day 181: number analyzed (Participants) | 198 | 257 | 269 | 59 | 85 | 83 | 74 | 57 | 51 | 66 | 25 | 25 | 116 | 68
  Day 181 | 20073 [17076 to 23596] | 20450 [18029 to 23195] | 18628 [16117 to 21530] | 25701 [17854 to 36998] | 25615 [20346 to 32248] | 24500 [19714 to 30448] | 7281 [5366 to 9880] | 8665 [6100 to 12311] | 10649 [7312 to 15510] | 12342 [8420 to 18092] | 11275 [7727 to 16451] | 19231 [12448 to 29712] | 21387 [17825 to 25661] | 20803 [16151 to 26794]
  Day 366: number analyzed (Participants) | 28 | 234 | 241 | 20 | 81 | 72 | 0 | 30 | 32 | 10 | 22 | 22 | 99 | 57
  Day 366 | 41232 [28233 to 60218] | 19545 [17037 to 22422] | 19989 [17351 to 23028] | 32368 [16026 to 65374] | 25800 [20031 to 33232] | 19848 [15543 to 25345] |  | 10382 [6531 to 16505] | 10937 [6565 to 18220] | 14545 [4542 to 46582] | 12176 [8897 to 16664] | 12002 [8266 to 17425] | 32168 [25602 to 40417] | 33194 [24774 to 44476]

11. Secondary Outcome: Phase 3: Cohorts 1 and 2: Number of Participants With >=2-Fold and >=4-Fold Rise in Binding Antibody Concentration Against SARS-CoV-2 D614G Strain at Days 15, 29, 91, 181, and 366
Description: as for outcome 5
Time Frame: Pre-vaccination on Day 1 and Post-vaccination on Days 15, 29, 91, 181, and 366
Population: The PPAS is a subset of the FAS. Only participants analyzed for each parameter at specific timepoint are reported. Results data was not collected for 'Phase 3-Exploratory reporting groups' because study vaccine used in exploratory arms were different from booster cohort. No participants were analyzed and thus data was not collected at Day 366 for "Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614)" reporting group.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351)
Number analyzed (Participants) | 312 | 332 | 340 | 106 | 98 | 101 | 119 | 94 | 93 | 96 | 34 | 34 | 124 | 72
Participants
  Day 15: >=2-fold rise: number analyzed (Participants) | 302 | 322 | 334 | 101 | 93 | 98 | 119 | 94 | 93 | 91 | 31 | 34 | 120 | 72
  Day 15: >=2-fold rise | 287 | 276 | 292 | 94 | 84 | 87 | 114 | 92 | 92 | 88 | 24 | 29 | 108 | 69
  Day 15: >=4-fold rise: number analyzed (Participants) | 302 | 322 | 334 | 101 | 93 | 98 | 119 | 94 | 93 | 91 | 31 | 34 | 120 | 72
  Day 15: >=4-fold rise | 265 | 234 | 265 | 72 | 73 | 69 | 106 | 85 | 90 | 84 | 19 | 28 | 103 | 67
  Day 29: >=2-fold rise: number analyzed (Participants) | 312 | 332 | 340 | 106 | 98 | 101 | 118 | 94 | 92 | 96 | 34 | 31 | 124 | 71
  Day 29: >=2-fold rise | 285 | 278 | 285 | 93 | 87 | 87 | 111 | 92 | 90 | 91 | 24 | 27 | 115 | 69
  Day 29: >=4-fold rise: number analyzed (Participants) | 312 | 332 | 340 | 106 | 98 | 101 | 118 | 94 | 92 | 96 | 34 | 31 | 124 | 71
  Day 29: >=4-fold rise | 253 | 243 | 254 | 71 | 75 | 74 | 96 | 85 | 86 | 84 | 19 | 27 | 109 | 66
  Day 91: >=2-fold rise: number analyzed (Participants) | 251 | 266 | 279 | 91 | 84 | 91 | 87 | 61 | 60 | 86 | 29 | 26 | 114 | 69
  Day 91: >=2-fold rise | 227 | 210 | 217 | 73 | 70 | 76 | 82 | 61 | 59 | 79 | 17 | 23 | 105 | 65
  Day 91: >=4-fold rise: number analyzed (Participants) | 251 | 266 | 279 | 91 | 84 | 91 | 87 | 61 | 60 | 86 | 29 | 26 | 114 | 69
  Day 91: >=4-fold rise | 197 | 183 | 184 | 60 | 62 | 58 | 69 | 57 | 56 | 72 | 14 | 22 | 98 | 62
  Day 181: >=2-fold rise: number analyzed (Participants) | 198 | 255 | 269 | 59 | 85 | 83 | 74 | 57 | 51 | 65 | 25 | 25 | 116 | 68
  Day 181: >=2-fold rise | 175 | 189 | 193 | 43 | 63 | 59 | 59 | 53 | 49 | 56 | 14 | 20 | 98 | 62
  Day 181: >=4-fold rise: number analyzed (Participants) | 198 | 255 | 269 | 59 | 85 | 83 | 74 | 57 | 51 | 65 | 25 | 25 | 116 | 68
  Day 181: >=4-fold rise | 146 | 160 | 167 | 38 | 55 | 48 | 45 | 45 | 40 | 51 | 11 | 17 | 89 | 59
  Day 366: >=2-fold rise: number analyzed (Participants) | 28 | 232 | 240 | 19 | 81 | 72 | 0 | 30 | 32 | 10 | 22 | 22 | 99 | 57
  Day 366: >=2-fold rise | 27 | 174 | 184 | 15 | 62 | 49 |  | 26 | 27 | 9 | 12 | 17 | 83 | 53
  Day 366: >=4-fold rise: number analyzed (Participants) | 28 | 232 | 240 | 19 | 81 | 72 | 0 | 30 | 32 | 10 | 22 | 22 | 99 | 57
  Day 366: >=4-fold rise | 26 | 147 | 165 | 13 | 56 | 37 |  | 23 | 23 | 7 | 11 | 14 | 77 | 52

12. Secondary Outcome: Phase 3: Cohort 2: Geometric Mean Titers of Neutralizing Antibodies Against SARS-CoV-2 D614G Strain and B.1.351 Variant at Days 1, 15, 29, and 91
Description: as for outcome 7
Time Frame: Pre-vaccination on Day 1 and post-vaccination on Days 15, 29, and 91
Population: The PPAS is a subset of the FAS. Only participants analyzed for each parameter at specific timepoint are reported. Results data was not collected for 'Phase 3-Exploratory reporting groups' because study vaccine used in exploratory arms were different from booster cohort.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351)
Number analyzed (Participants) | 348 | 345 | 107 | 101 | 94 | 97 | 36 | 36 | 123 | 72
titers
  Day 1: D614G: number analyzed (Participants) | 348 | 345 | 107 | 101 | 89 | 93 | 36 | 36 | 107 | 67
  Day 1: D614G | 678 [558 to 824] | 579 [478 to 701] | 1107 [816 to 1503] | 1347 [977 to 1858] | 137 [98.0 to 193] | 134 [95.7 to 186] | 1188 [567 to 2490] | 447 [217 to 921] | 274 [182 to 413] | 159 [97.4 to 260]
  Day 1: B.1.351: number analyzed (Participants) | 336 | 324 | 97 | 94 | 90 | 97 | 36 | 34 | 108 | 68
  Day 1: B.1.351 | 176 [142 to 217] | 149 [120 to 184] | 258 [182 to 364] | 296 [207 to 424] | 43.3 [32.0 to 58.5] | 36.8 [28.8 to 47.1] | 345 [167 to 714] | 122 [55.3 to 268] | 97.7 [68.0 to 140] | 70.3 [47.9 to 103]
  Day 15: D614G: number analyzed (Participants) | 325 | 334 | 93 | 96 | 94 | 93 | 31 | 34 | 119 | 72
  Day 15: D614G | 9995 [8976 to 11129] | 8430 [7572 to 9386] | 14240 [11257 to 18013] | 12522 [10368 to 15123] | 5536 [4436 to 6910] | 5855 [4669 to 7344] | 11005 [7533 to 16078] | 11624 [8086 to 16710] | 22457 [19123 to 26374] | 25002 [18441 to 33897]
  Day 15: B.1.351: number analyzed (Participants) | 325 | 334 | 93 | 95 | 94 | 93 | 30 | 34 | 119 | 72
  Day 15: B.1.351 | 7021 [6262 to 7873] | 4900 [4370 to 5494] | 9449 [7376 to 12104] | 6581 [5340 to 8111] | 4610 [3689 to 5760] | 3099 [2386 to 4026] | 6872 [4482 to 10537] | 5057 [3416 to 7488] | 7452 [6212 to 8939] | 13300 [9817 to 18018]
  Day 29: D614G: number analyzed (Participants) | 333 | 341 | 99 | 100 | 93 | 92 | 34 | 31 | 123 | 71
  Day 29: D614G | 14065 [12399 to 15954] | 10885 [9664 to 12261] | 16286 [12808 to 20710] | 16874 [13763 to 20688] | 6320 [4941 to 8083] | 6370 [5014 to 8093] | 9711 [6526 to 14450] | 9521 [6555 to 13828] | 16032 [13535 to 18989] | 16425 [12103 to 22291]
  Day 29: B.1.351: number analyzed (Participants) | 333 | 340 | 99 | 98 | 93 | 92 | 34 | 31 | 123 | 71
  Day 29: B.1.351 | 8947 [7845 to 10203] | 6045 [5307 to 6886] | 10264 [7924 to 13296] | 8139 [6470 to 10239] | 4736 [3680 to 6096] | 3103 [2340 to 4115] | 6028 [3889 to 9342] | 4007 [2553 to 6290] | 7185 [5841 to 8838] | 12712 [9376 to 17234]
  Day 91: D614G: number analyzed (Participants) | 264 | 279 | 84 | 89 | 61 | 60 | 29 | 26 | 112 | 69
  Day 91: D614G | 11037 [9530 to 12782] | 8523 [7284 to 9973] | 13701 [10206 to 18392] | 12424 [9586 to 16103] | 3620 [2680 to 4891] | 3981 [2812 to 5637] | 5797 [3725 to 9024] | 5880 [3125 to 11064] | 14498 [11931 to 17618] | 13641 [9766 to 19055]
  Day 91: B.1.351: number analyzed (Participants) | 264 | 279 | 84 | 89 | 61 | 60 | 29 | 26 | 112 | 69
  Day 91: B.1.351 | 6557 [5617 to 7654] | 4359 [3673 to 5172] | 8141 [5982 to 11080] | 5474 [4176 to 7175] | 2456 [1792 to 3364] | 2029 [1376 to 2993] | 3374 [2161 to 5269] | 2405 [1093 to 5295] | 6455 [5117 to 8143] | 8990 [6284 to 12861]

13. Secondary Outcome: Phase 3: Cohort 2: Number of Participants With >=2-Fold and >=4-Fold Rise in Serum Neutralization Antibody Titers Against SARS-CoV-2 D614G Strain and B.1.351 Variant at Days 15, 29, and 91
Description: as for outcome 8
Time Frame: Pre-vaccination on Day 1 and Post-vaccination on Days 15, 29, and 91
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351)
Number analyzed (Participants) | 318 | 324 | 99 | 95 | 87 | 91 | 33 | 33 | 103 | 64
Participants
  D614G; Day 15: >=2-fold rise: number analyzed (Participants) | 315 | 320 | 92 | 91 | 87 | 88 | 31 | 33 | 99 | 64
  D614G; Day 15: >=2-fold rise | 267 | 269 | 79 | 77 | 85 | 84 | 26 | 30 | 86 | 60
  D614G; Day 15: >=4-fold rise: number analyzed (Participants) | 315 | 320 | 92 | 91 | 87 | 88 | 31 | 33 | 99 | 64
  D614G; Day 15: >=4-fold rise | 232 | 242 | 67 | 58 | 78 | 79 | 18 | 26 | 84 | 58
  D614G; Day 29: >=2-fold rise: number analyzed (Participants) | 318 | 324 | 99 | 95 | 86 | 86 | 33 | 30 | 101 | 62
  D614G; Day 29: >=2-fold rise | 272 | 283 | 83 | 76 | 84 | 83 | 22 | 28 | 89 | 58
  D614G; Day 29: >=4-fold rise: number analyzed (Participants) | 318 | 324 | 99 | 95 | 86 | 86 | 33 | 30 | 101 | 62
  D614G; Day 29: >=4-fold rise | 240 | 251 | 74 | 67 | 80 | 80 | 15 | 23 | 85 | 56
  D614G; Day 91: >=2-fold rise: number analyzed (Participants) | 251 | 265 | 84 | 86 | 58 | 55 | 28 | 25 | 93 | 61
  D614G; Day 91: >=2-fold rise | 199 | 208 | 69 | 70 | 57 | 51 | 16 | 20 | 81 | 57
  D614G; Day 91: >=4-fold rise: number analyzed (Participants) | 251 | 265 | 84 | 86 | 58 | 55 | 28 | 25 | 93 | 61
  D614G; Day 91: >=4-fold rise | 175 | 187 | 57 | 54 | 55 | 48 | 12 | 16 | 78 | 53
  B.1.351; Day 15: >=2-fold rise: number analyzed (Participants) | 299 | 298 | 84 | 85 | 87 | 91 | 29 | 31 | 99 | 64
  B.1.351; Day 15: >=2-fold rise | 275 | 269 | 77 | 79 | 85 | 88 | 28 | 28 | 88 | 62
  B.1.351; Day 15: >=4-fold rise: number analyzed (Participants) | 299 | 298 | 84 | 85 | 87 | 91 | 29 | 31 | 99 | 64
  B.1.351; Day 15: >=4-fold rise | 249 | 247 | 70 | 68 | 83 | 88 | 22 | 24 | 85 | 58
  B.1.351; Day 29: >=2-fold rise: number analyzed (Participants) | 306 | 304 | 90 | 88 | 87 | 90 | 33 | 28 | 103 | 64
  B.1.351; Day 29: >=2-fold rise | 278 | 277 | 81 | 79 | 86 | 87 | 28 | 26 | 95 | 62
  B.1.351; Day 29: >=4-fold rise: number analyzed (Participants) | 306 | 304 | 90 | 88 | 87 | 90 | 33 | 28 | 103 | 64
  B.1.351; Day 29: >=4-fold rise | 258 | 261 | 75 | 70 | 84 | 87 | 20 | 25 | 92 | 58
  B.1.351; Day 91: >=2-fold rise: number analyzed (Participants) | 246 | 252 | 76 | 82 | 56 | 58 | 29 | 25 | 94 | 62
  B.1.351; Day 91: >=2-fold rise | 212 | 207 | 69 | 68 | 56 | 56 | 22 | 21 | 87 | 58
  B.1.351; Day 91: >=4-fold rise: number analyzed (Participants) | 246 | 252 | 76 | 82 | 56 | 58 | 29 | 25 | 94 | 62
  B.1.351; Day 91: >=4-fold rise | 195 | 197 | 62 | 60 | 56 | 53 | 16 | 17 | 80 | 55

14. Secondary Outcome: Phase 3: Comparator: Geometric Mean Titers of Neutralizing Antibodies Against SARS-CoV-2 D614G Strain and B.1.351 Variant at Days 1, 22, 36, 134, 202, 292, and 387
Description: as for outcome 7
Time Frame: Pre-vaccination on Day 1 and post-vaccination on Days 22, 36, 134, 202, 292, and 387
Population: The PPAS is a subset of the FAS. Only participants analyzed for each parameter at specific timepoint are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614)
Number analyzed (Participants) | 330
titers
  D614G: Day 1 | 20.3 [19.7 to 21.0]
  D614G: Day 22: number analyzed (Participants) | 281
  D614G: Day 22 | 53.3 [44.6 to 63.8]
  D614G: Day 36: number analyzed (Participants) | 302
  D614G: Day 36 | 3658 [3123 to 4286]
  D614G: Day 134: number analyzed (Participants) | 143
  D614G: Day 134 | 1050 [743 to 1486]
  D614G: Day 202: number analyzed (Participants) | 128
  D614G: Day 202 | 1685 [1142 to 2487]
  D614G: Day 292: number analyzed (Participants) | 117
  D614G: Day 292 | 1943 [1294 to 2918]
  D614G: Day 387: number analyzed (Participants) | 112
  D614G: Day 387 | 1973 [1344 to 2897]
  B.1.351: Day 1: number analyzed (Participants) | 329
  B.1.351: Day 1 | 20.3 [19.7 to 20.8]
  B.1.351: Day 22: number analyzed (Participants) | 326
  B.1.351: Day 22 | 29.4 [25.7 to 33.5]
  B.1.351: Day 36: number analyzed (Participants) | 291
  B.1.351: Day 36 | 413 [346 to 493]
  B.1.351: Day 134: number analyzed (Participants) | 113
  B.1.351: Day 134 | 496 [330 to 745]
  B.1.351: Day 202: number analyzed (Participants) | 123
  B.1.351: Day 202 | 671 [441 to 1022]
  B.1.351: Day 292: number analyzed (Participants) | 120
  B.1.351: Day 292 | 867 [560 to 1342]
  B.1.351: Day 387: number analyzed (Participants) | 112
  B.1.351: Day 387 | 1033 [686 to 1555]

15. Secondary Outcome: Phase 3: Comparator: Number of Participants With >=2-Fold and >=4-Fold Rise in Serum Neutralization Antibody Titers Against SARS-CoV-2 D614G Strain and B.1.351 Variant at Days 22, 36, 134, 202, 292, and 387
Description: as for outcome 8
Time Frame: Pre-vaccination on Day 1 and Post-vaccination on Days 22, 36, 134, 202, 292, and 387
Population: The PPAS is a subset of the FAS. Only participants analyzed for each parameter at specific timepoint are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614)
Number analyzed (Participants) | 325
Participants
  D614G; Day 22: >=2-fold rise: number analyzed (Participants) | 281
  D614G; Day 22: >=2-fold rise | 99
  D614G; Day 22: >=4-fold rise: number analyzed (Participants) | 281
  D614G; Day 22: >=4-fold rise | 88
  D614G; Day 36: >=2-fold rise: number analyzed (Participants) | 301
  D614G; Day 36: >=2-fold rise | 299
  D614G; Day 36: >=4-fold rise: number analyzed (Participants) | 301
  D614G; Day 36: >=4-fold rise | 298
  D614G; Day 134: >=2-fold rise: number analyzed (Participants) | 143
  D614G; Day 134: >=2-fold rise | 134
  D614G; Day 134: >=4-fold rise: number analyzed (Participants) | 143
  D614G; Day 134: >=4-fold rise | 131
  D614G; Day 202: >=2-fold rise: number analyzed (Participants) | 127
  D614G; Day 202: >=2-fold rise | 120
  D614G; Day 202: >=4-fold rise: number analyzed (Participants) | 127
  D614G; Day 202: >=4-fold rise | 119
  D614G; Day 292: >=2-fold rise: number analyzed (Participants) | 117
  D614G; Day 292: >=2-fold rise | 108
  D614G; Day 292: >=4-fold rise: number analyzed (Participants) | 117
  D614G; Day 292: >=4-fold rise | 105
  D614G; Day 387: >=2-fold rise: number analyzed (Participants) | 111
  D614G; Day 387: >=2-fold rise | 105
  D614G; Day 387: >=4-fold rise: number analyzed (Participants) | 111
  D614G; Day 387: >=4-fold rise | 101
  B.1.351; Day 22: >=2-fold rise | 39
  B.1.351; Day 22: >=4-fold rise | 32
  B.1.351; Day 36: >=2-fold rise: number analyzed (Participants) | 290
  B.1.351; Day 36: >=2-fold rise | 264
  B.1.351; Day 36: >=4-fold rise: number analyzed (Participants) | 290
  B.1.351; Day 36: >=4-fold rise | 251
  B.1.351; Day 134: >=2-fold rise: number analyzed (Participants) | 112
  B.1.351; Day 134: >=2-fold rise | 99
  B.1.351; Day 134: >=4-fold rise: number analyzed (Participants) | 112
  B.1.351; Day 134: >=4-fold rise | 89
  B.1.351; Day 202: >=2-fold rise: number analyzed (Participants) | 122
  B.1.351; Day 202: >=2-fold rise | 100
  B.1.351; Day 202: >=4-fold rise: number analyzed (Participants) | 122
  B.1.351; Day 202: >=4-fold rise | 97
  B.1.351; Day 292: >=2-fold rise: number analyzed (Participants) | 119
  B.1.351; Day 292: >=2-fold rise | 98
  B.1.351; Day 292: >=4-fold rise: number analyzed (Participants) | 119
  B.1.351; Day 292: >=4-fold rise | 91
  B.1.351; Day 387: >=2-fold rise: number analyzed (Participants) | 111
  B.1.351; Day 387: >=2-fold rise | 96
  B.1.351; Day 387: >=4-fold rise: number analyzed (Participants) | 111
  B.1.351; Day 387: >=4-fold rise | 94

16. Secondary Outcome: Phase 3: Comparator: Geometric Mean Concentration of Binding Antibodies Against SARS-CoV-2 D614G Strain at Days 1, 22, 36, 134, 202, 292, and 387
Description: as for outcome 10
Time Frame: Pre-vaccination on Day 1 and post-vaccination on Days 22, 36, 134, 202, 292, and 387
Population: The PPAS is a subset of the FAS. Only participants analyzed at specific timepoint are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614)
Number analyzed (Participants) | 330
titers
  Day 1: number analyzed (Participants) | 326
  Day 1 | 10.7 [9.91 to 11.6]
  Day 22 | 212 [183 to 246]
  Day 36: number analyzed (Participants) | 303
  Day 36 | 24278 [21681 to 27185]
  Day 134: number analyzed (Participants) | 147
  Day 134 | 6593 [4952 to 8779]
  Day 202: number analyzed (Participants) | 132
  Day 202 | 6667 [4833 to 9197]
  Day 292: number analyzed (Participants) | 122
  Day 292 | 6868 [4919 to 9587]
  Day 387: number analyzed (Participants) | 115
  Day 387 | 7112 [5216 to 9697]

17. Secondary Outcome: Phase 3: Comparator: Number of Participants With >=2-Fold and >=4-Fold Rise in Binding Antibody Concentration Against SARS-CoV-2 D614G Strain at Days 22, 36, 134, 202, 292, and 387
Description: as for outcome 5
Time Frame: Pre-vaccination on Day 1 and Post-vaccination on Days 22, 36, 134, 202, 292, and 387
Population: The PPAS is a subset of the FAS. Only participants analyzed for each parameter at specific timepoint are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614)
Number analyzed (Participants) | 331
Participants
  Day 22: >=2-fold rise | 312
  Day 22: >=4-fold rise | 290
  Day 36: >=2-fold rise: number analyzed (Participants) | 303
  Day 36: >=2-fold rise | 302
  Day 36: >=4-fold rise: number analyzed (Participants) | 303
  Day 36: >=4-fold rise | 302
  Day 134: >=2-fold rise: number analyzed (Participants) | 150
  Day 134: >=2-fold rise | 149
  Day 134: >=4-fold rise: number analyzed (Participants) | 150
  Day 134: >=4-fold rise | 148
  Day 202: >=2-fold rise: number analyzed (Participants) | 134
  Day 202: >=2-fold rise | 133
  Day 202: >=4-fold rise: number analyzed (Participants) | 134
  Day 202: >=4-fold rise | 133
  Day 292: >=2-fold rise: number analyzed (Participants) | 124
  Day 292: >=2-fold rise | 123
  Day 292: >=4-fold rise: number analyzed (Participants) | 124
  Day 292: >=4-fold rise | 123
  Day 387: >=2-fold rise: number analyzed (Participants) | 118
  Day 387: >=2-fold rise | 117
  Day 387: >=4-fold rise: number analyzed (Participants) | 118
  Day 387: >=4-fold rise | 117

18. Secondary Outcome: Phase 3: Comparator: Percentage of Responders as Determined by Binding Antibody Concentration Against SARS-CoV-2 D614G Strain at Days 22, 36, 134, 202, 292, and 387
Description: Responders were participants who had baseline values below LLOQ with detectable antibody concentration above assay LLOQ at each pre-defined post-vaccination time point and participants with baseline values above LLOQ with a 4-fold increase in neutralizing antibody titers at each pre-defined post-vaccination time point. Binding antibodies activity against SARS-CoV-2 D614G strain was measured with Nexelis GCN4 S-ELISA. Percentages are rounded off to the tenth decimal place.
Time Frame: Post-vaccination on Days 22, 36, 134, 202, 292, and 387
Population: The PPAS is a subset of the FAS. Only participants analyzed at specific timepoint are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614)
Number analyzed (Participants) | 331
percentage of participants
  Day 22 | 94.3 [91.2 to 96.5]
  Day 36: number analyzed (Participants) | 325
  Day 36 | 99.7 [98.3 to 100]
  Day 134: number analyzed (Participants) | 159
  Day 134 | 98.7 [95.5 to 99.8]
  Day 202: number analyzed (Participants) | 141
  Day 202 | 99.3 [96.1 to 100]
  Day 292: number analyzed (Participants) | 134
  Day 292 | 99.3 [95.9 to 100]
  Day 387: number analyzed (Participants) | 127
  Day 387 | 99.2 [95.7 to 100]

19. Secondary Outcome: Phase 2: Percentage of Participants With Serologically-Confirmed SARS-CoV-2 Infection
Description: Blood samples collected from participants were used for serological assessments in the study. Serologically-confirmed SARS-CoV-2 infection was defined as a positive result in a serum sample for antibodies specific to the nucleocapsid of SARS-CoV-2 detected by electrochemiluminescence immunoassay. Percentages are rounded off to the tenth decimal place.
Time Frame: From first dose of study vaccine administration (Day 1) up to 387 days
Population: The Safety analysis set included participants randomized and who had received at least 1 dose of the study vaccines. One participant from "Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3" received the vaccine formulation of "Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2". So, number of participants analyzed was 240 (N) for "Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2".
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3
Number analyzed (Participants) | 240 | 240 | 241
percentage of participants | 12.1 [8.2 to 16.9] | 10.8 [7.2 to 15.5] | 14.1 [10.0 to 19.2]

20. Secondary Outcome: Phase 2 and Phase 3 (Cohorts 1, 2 and Comparator): Percentage of Participants With Laboratory-Confirmed Symptomatic COVID-19
Description: Laboratory-confirmed SARS-CoV-2 infection was defined as a positive result for SARS-CoV-2 by nucleic acid amplification test (done by the central laboratory or locally) on at least 1 respiratory sample. Percentages are rounded off to the tenth decimal place.
Time Frame: Phase 2 and Phase 3 Comparator: From first dose of study vaccine administration (Day 1) up to 387 days. Phase 3 Cohorts 1 and 2: From first dose of study vaccine administration (Day 1) up to 366 days.
Population: Safety analysis set included participants randomized and who had received at least 1 dose of study vaccines. 1 participant from "Phase 2:CoV2 preS dTM-AS03(D614) Formulation 3" received vaccine formulation of "Phase 2:CoV2 preS dTM-AS03(D614) Formulation 2". So, number analyzed was 240(N) for "Phase 2:CoV2 preS dTM-AS03(D614) Formulation 2". Results data was not collected for 'Phase 3-Exploratory reporting groups' because study vaccine used in exploratory arms were different from booster cohort.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3 | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614)
Number analyzed (Participants) | 240 | 240 | 241 | 328 | 378 | 375 | 113 | 111 | 108 | 127 | 100 | 100 | 103 | 38 | 38 | 132 | 78 | 473
percentage of participants | 3.3 [1.4 to 6.5] | 1.7 [0.5 to 4.2] | 5.4 [2.9 to 9.0] | 14.0 [10.5 to 18.3] | 20.9 [16.9 to 25.4] | 23.5 [19.3 to 28.1] | 12.4 [6.9 to 19.9] | 10.8 [5.7 to 18.1] | 10.2 [5.2 to 17.5] | 24.4 [17.2 to 32.8] | 25.0 [16.9 to 34.7] | 29.0 [20.4 to 38.9] | 9.7 [4.8 to 17.1] | 0 [0 to 9.3] | 18.4 [7.7 to 34.3] | 18.9 [12.6 to 26.7] | 19.2 [11.2 to 29.7] | 8.2 [5.9 to 11.1]

21. Secondary Outcome: Phase 2 and Phase 3 (Cohorts 1, 2 and Comparator): Percentage of Participants With Symptomatic COVID-19 Episodes Associated With Hospitalization
Description: Symptomatic COVID-19 was defined as laboratory-confirmed SARS-CoV-2 infection accompanied by protocol-defined COVID-19-like illness. Percentages are rounded off to the tenth decimal place.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3 | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614)
Number analyzed (Participants) | 240 | 240 | 241 | 328 | 378 | 375 | 113 | 111 | 108 | 127 | 100 | 100 | 103 | 38 | 38 | 132 | 78 | 473
percentage of participants | 0 [0 to 1.5] | 0 [0 to 1.5] | 0 [0 to 1.5] | 0 [0 to 1.1] | 0 [0 to 1.0] | 0.3 [0 to 1.5] | 0 [0 to 3.2] | 0 [0 to 3.3] | 0 [0 to 3.4] | 0.8 [0 to 4.3] | 0 [0 to 3.6] | 0 [0 to 3.6] | 0 [0 to 3.5] | 0 [0 to 9.3] | 0 [0 to 9.3] | 0 [0 to 2.8] | 0 [0 to 4.6] | 0 [0 to 0.8]

22. Secondary Outcome: Phase 2 and Phase 3 (Cohorts 1, 2 and Comparator): Percentage of Participants With Severe Symptomatic COVID-19
Description: Severe COVID-19 was defined as COVID-19 with any 1: Any clinical signs of severe illness measured at least on 2 occasions separated by 30 minutes, supplemental oxygen administration for >1 hour, use of invasive or non-invasive ventilation or Extracorporeal Membrane Oxygenation, clinical diagnosis of respiratory failure, significant acute renal, hepatic, or neurologic dysfunction, shock (defined by systolic blood pressure ˂90 millimeter of mercury (mmHg), or diastolic blood pressure ˂60 mmHg or requiring vasopressors), admission to an intensive care unit, or death. Symptomatic COVID-19 was defined as laboratory-confirmed SARS-CoV-2 infection accompanied by protocol-defined COVID-19-like illness. Percentages are rounded off to the tenth decimal place.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3 | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614)
Number analyzed (Participants) | 240 | 240 | 241 | 328 | 378 | 375 | 113 | 111 | 108 | 127 | 100 | 100 | 103 | 38 | 38 | 132 | 78 | 473
percentage of participants | 0 [0 to 1.5] | 0 [0 to 1.5] | 0 [0 to 1.5] | 0 [0 to 1.1] | 0 [0 to 1.0] | 0.3 [0 to 1.5] | 0 [0 to 3.2] | 0 [0 to 3.3] | 0 [0 to 3.4] | 0 [0 to 2.9] | 0 [0 to 3.6] | 0 [0 to 3.6] | 0 [0 to 3.5] | 0 [0 to 9.3] | 0 [0 to 9.3] | 0.8 [0 to 4.1] | 0 [0 to 4.6] | 0 [0 to 0.8]

23. Secondary Outcome: Phase 2 and Phase 3 (Cohorts 1, 2 and Comparator): Percentage of Participants With Death Associated With Symptomatic COVID-19
Description: Death associated with COVID-19 was defined as death in a participant with COVID-19 who died within 28 days of the first positive specimen date OR died more than 28 days after the first specimen date and COVID-19 was mentioned as an immediate or underlying cause of death on the death certificate. Symptomatic COVID-19 was defined as laboratory-confirmed SARS-CoV-2 infection accompanied by protocol-defined COVID-19-like illness. Percentages are rounded off to the tenth decimal place.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3 | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614)
Number analyzed (Participants) | 240 | 240 | 241 | 328 | 378 | 375 | 113 | 111 | 108 | 127 | 100 | 100 | 103 | 38 | 38 | 132 | 78 | 473
percentage of participants | 0 [0 to 1.5] | 0 [0 to 1.5] | 0 [0 to 1.5] | 0 [0 to 1.1] | 0 [0 to 1.0] | 0 [0 to 1.0] | 0 [0 to 3.2] | 0 [0 to 3.3] | 0 [0 to 3.4] | 0 [0 to 2.9] | 0 [0 to 3.6] | 0 [0 to 3.6] | 0 [0 to 3.5] | 0 [0 to 9.3] | 0 [0 to 9.3] | 0 [0 to 2.8] | 0 [0 to 4.6] | 0 [0 to 0.8]

24. Primary Outcome: Phase 2 and Phase 3 (Cohorts 1, 2 and Comparator): Number of Participants With Immediate Unsolicited Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Immediate events were recorded to capture medically relevant unsolicited systemic AEs which occurred within the first 30 minutes after vaccination. An unsolicited AE was an observed AE that did not fulfill the conditions of solicited reactions, that is, pre-listed in the case report form (CRF) in terms of diagnosis and onset window post-vaccination.
Time Frame: Up to 30 minutes after each vaccination (Phase 2: Postdose on Days 1 and 22; Phase 3: Between 4 to 10 months after priming vaccine)
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3 | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614)
Number analyzed (Participants) | 240 | 240 | 241 | 328 | 378 | 375 | 113 | 111 | 108 | 127 | 100 | 100 | 103 | 38 | 38 | 132 | 78 | 473
Participants | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9

25. Primary Outcome: Phase 2 and Phase 3 (Cohorts 1, 2 and Comparator): Number of Participants With Solicited Injection Site Reactions and Systemic Reactions
Description: A solicited reaction was an "expected" adverse reaction (AR) (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRF, and were considered to be related to the study vaccine administered. An injection site reaction was an AR at and around the injection site of the study vaccine. Systemic AR were all ARs that were not injection site reactions.
Time Frame: Up to 7 days after each vaccination (Phase 2: Postdose on Days 1 and 22; Phase 3: Between 4 to 10 months after priming vaccine)
Population: The Safety analysis set included participants randomized and who had received at least 1 dose of the study vaccines. Safety analysis was performed according to the actual study vaccine received by the participants. Results data was not collected for 'Phase 3-Exploratory reporting groups' because study vaccine used in exploratory arms were different from booster cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3 | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614)
Number analyzed (Participants) | 238 | 237 | 239 | 326 | 367 | 370 | 113 | 110 | 108 | 127 | 100 | 100 | 102 | 38 | 38 | 132 | 78 | 460
Participants
  Injection site reaction | 201 | 196 | 200 | 262 | 300 | 303 | 90 | 82 | 74 | 104 | 87 | 87 | 81 | 19 | 19 | 98 | 46 | 375
  Systemic reaction | 191 | 191 | 185 | 198 | 238 | 242 | 67 | 67 | 65 | 75 | 61 | 75 | 62 | 14 | 17 | 88 | 36 | 359

26. Primary Outcome: Phase 2 and Phase 3 (Cohorts 1, 2 and Comparator): Number of Participants With Unsolicited Adverse Events
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An unsolicited AE was an observed AE that did not fulfill the conditions of solicited reactions, that is, pre-listed in the CRF in terms of diagnosis and onset window post-vaccination.
Time Frame: Up to 21 days after each vaccination (Phase 2: Postdose on Days 1 and 22; Phase 3: Between 4 to 10 months after priming vaccine)
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3 | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614)
Number analyzed (Participants) | 240 | 240 | 241 | 328 | 378 | 375 | 113 | 111 | 108 | 127 | 100 | 100 | 103 | 38 | 38 | 132 | 78 | 473
Participants | 88 | 81 | 91 | 76 | 106 | 96 | 29 | 18 | 22 | 34 | 27 | 35 | 16 | 7 | 7 | 25 | 11 | 199

27. Primary Outcome: Phase 2 and Phase 3 (Cohorts 1, 2 and Comparator): Number of Participants With Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs) and Medically Attended Adverse Events (MAAEs)
Description: An SAE was defined as any AE that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. An AESI (serious or non-serious) was 1 of scientific and medical concern specific to the Sponsor's study intervention or program, for which ongoing monitoring and rapid communication by the Investigator to the Sponsor could be appropriate. An MAAE was a new onset or a worsening of a condition that prompted the participant or participant's parent/guardian to seek unplanned medical advice at a physician's office or Emergency Department.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3 | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614)
Number analyzed (Participants) | 240 | 240 | 241 | 328 | 378 | 375 | 113 | 111 | 108 | 127 | 100 | 100 | 103 | 38 | 38 | 132 | 78 | 473
Participants
  SAE | 2 | 6 | 4 | 8 | 9 | 11 | 3 | 1 | 4 | 3 | 4 | 0 | 1 | 2 | 3 | 3 | 3 | 14
  AESI | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  MAAE | 42 | 48 | 59 | 80 | 106 | 117 | 28 | 25 | 19 | 31 | 24 | 29 | 19 | 7 | 7 | 42 | 32 | 110

28. Primary Outcome: Phase 2: Geometric Mean Titers (GMTs) of Neutralizing Antibodies Against Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV-2) D614G Strain at Day 1
Description: as for outcome 1
Time Frame: Pre-vaccination on Day 1
Population: The per-protocol analysis set (PPAS) Naïve-D01+D22 is a subset of the full analysis set (FAS).
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3
Number analyzed (Participants) | 167 | 170 | 171
titers | 20.0 [NA to NA] — Since all participants have 20 titers at Day 1, leading to a zero standard error, this makes it impossible to calculate a meaningful confidence interval. | 20.0 [NA to NA] — Since all participants have 20 titers at Day 1, leading to a zero standard error, this makes it impossible to calculate a meaningful confidence interval. | 20.0 [NA to NA] — Since all participants have 20 titers at Day 1, leading to a zero standard error, this makes it impossible to calculate a meaningful confidence interval.

29. Primary Outcome: Phase 2: Geometric Mean Titers of Neutralizing Antibodies Against SARS-CoV-2 D614G Strain at Day 36
Description: as for outcome 1
Time Frame: Day 36
Population: The PPAS Naïve-D01+D22 is a subset of the FAS. Only participants analyzed at Day 36 are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3
Number analyzed (Participants) | 162 | 163 | 167
titers | 2132 [1690 to 2688] | 2376 [1873 to 3015] | 2903 [2289 to 3683]

30. Primary Outcome: Phase 2: Number of Participants With >=2-Fold and >=4-Fold Rise in Serum Neutralization Antibody Titers Against SARS-CoV-2 D614G Strain at Day 36
Description: as for outcome 2
Time Frame: Day 1 (pre-vaccination) and Day 36
Population: The PPAS Naïve-D01+D22 is a subset of the FAS. Only participants analyzed at specific timepoint are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3
Number analyzed (Participants) | 159 | 158 | 161
Participants
  >=2-fold rise | 155 | 156 | 158
  >=4-fold rise | 154 | 154 | 157

31. Primary Outcome: Phase 2: Number of Responders as Determined by Neutralizing Antibody Titers Against SARS-CoV-2 D614G Strain at Day 36
Description: Responders were participants who had baseline values below lower limit of quantification (LLOQ) with detectable neutralization titer above assay LLOQ at each pre-defined post-vaccination time point and participants with baseline values above LLOQ with a 4-fold increase in neutralizing antibody titers at each pre-defined post-vaccination time point.
Time Frame: Day 36
Population: The PPAS Naïve-D01+D22 is a subset of the FAS. Only participants analyzed at Day 36 are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3
Number analyzed (Participants) | 159 | 158 | 161
Participants | 155 | 156 | 158

32. Primary Outcome: Phase 3: Cohorts 1 and 2: Geometric Mean Titers of Neutralizing Antibodies Against SARS-CoV-2 D614G Strain and B.1.351 Variant at Day 1
Description: as for outcome 7
Time Frame: Pre-vaccination on Day 1
Population: The PPAS is a subset of the FAS. Only participants analyzed for each parameter are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351)
Number analyzed (Participants) | 301 | 348 | 345 | 107 | 107 | 101 | 120 | 90 | 97 | 89 | 36 | 36 | 108 | 68
titers
  D614G: number analyzed (Participants) | 301 | 348 | 345 | 107 | 107 | 101 | 107 | 89 | 93 | 82 | 36 | 36 | 107 | 67
  D614G | 320 [275 to 373] | 678 [558 to 824] | 579 [478 to 701] | 668 [537 to 830] | 1107 [816 to 1503] | 1347 [977 to 1858] | 265 [190 to 369] | 137 [98.0 to 193] | 134 [95.7 to 186] | 222 [155 to 318] | 1188 [567 to 2490] | 447 [217 to 921] | 274 [182 to 413] | 159 [97.4 to 260]
  B.1.351: number analyzed (Participants) | 290 | 336 | 324 | 88 | 97 | 94 | 120 | 90 | 97 | 89 | 36 | 34 | 108 | 68
  B.1.351 | 70.1 [60.3 to 81.4] | 176 [142 to 217] | 149 [120 to 184] | 122 [95.4 to 157] | 258 [182 to 364] | 296 [207 to 424] | 54.1 [41.4 to 70.7] | 43.3 [32.0 to 58.5] | 36.8 [28.8 to 47.1] | 42.6 [32.5 to 55.7] | 345 [167 to 714] | 122 [55.3 to 268] | 97.7 [68.0 to 140] | 70.3 [47.9 to 103]

33. Primary Outcome: Phase 3: Cohorts 1, 2 and Comparator: Geometric Mean Titers of Neutralizing Antibodies Against SARS-CoV-2 D614G Strain and B.1.351 Variant at 14 Days Post-Vaccination
Description: as for outcome 7
Time Frame: Cohorts 1 and 2: 14 days post-vaccination on Day 1, Day 15; Comparator: 14 days post-vaccination on Day 22, Day 36
Population: The PPAS is a subset of the FAS. Only participants analyzed for each parameter are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614)
Number analyzed (Participants) | 301 | 325 | 334 | 101 | 93 | 96 | 118 | 94 | 93 | 91 | 31 | 34 | 119 | 72 | 307
titers
  D614G | 6964 [6268 to 7737] | 9995 [8976 to 11129] | 8430 [7572 to 9386] | 6347 [5207 to 7736] | 14240 [11257 to 18013] | 12522 [10368 to 15123] | 6257 [5313 to 7369] | 5536 [4436 to 6910] | 5855 [4669 to 7344] | 6875 [5587 to 8460] | 11005 [7533 to 16078] | 11624 [8086 to 16710] | 22457 [19123 to 26374] | 25002 [18441 to 33897] | 3611 [3086 to 4224]
  B.1.351: number analyzed (Participants) | 299 | 325 | 334 | 98 | 93 | 95 | 118 | 94 | 93 | 89 | 30 | 34 | 119 | 72 | 296
  B.1.351 | 2610 [2316 to 2942] | 7021 [6262 to 7873] | 4900 [4370 to 5494] | 2222 [1754 to 2814] | 9449 [7376 to 12104] | 6581 [5340 to 8111] | 2062 [1708 to 2489] | 4610 [3689 to 5760] | 3099 [2386 to 4026] | 2054 [1642 to 2568] | 6872 [4482 to 10537] | 5057 [3416 to 7488] | 7452 [6212 to 8939] | 13300 [9817 to 18018] | 413 [346 to 493]

34. Primary Outcome: Phase 3: Comparator: Percentage of Responders as Determined by Neutralizing Antibody Titers Against SARS-CoV-2 D614G Strain and B.1.351 Variant at Day 36
Description: Responders were participants who had baseline values below LLOQ with detectable neutralization titer above assay LLOQ at each pre-defined post-vaccination time point and participants with baseline values above LLOQ with a 4-fold increase in neutralizing antibody titers at each pre-defined post-vaccination time point. Percentages are rounded off to the tenth decimal place.
Time Frame: Day 36
Population: The PPAS is a subset of the FAS. Only participants analyzed for each parameter are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614)
Number analyzed (Participants) | 301
percentage of participants
  D614G | 99.3 [97.6 to 99.9]
  B.1.351: number analyzed (Participants) | 290
  B.1.351 | 91.0 [87.1 to 94.1]

ADVERSE EVENTS:
Time Frame: Phase 2 and Phase 3 Comparator: AEs data was collected from first dose of study vaccine administration (Day 1) up to 387 days. Phase 3 Cohorts 1 and 2: AEs data was collected from first dose of study vaccine administration (Day 1) up to 366 days.
Description: Analysis was performed on the safety analysis set. Safety analysis was performed according to the actual study vaccine received by the participants. One participant from "Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3" received the vaccine formulation of "Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2". So, number of participants analyzed was 240 (N) for "Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2".
Arm/Group | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3 | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351) | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614) | Phase 3: Exploratory 1: PBP - CoV2 preS dTM (B.1.351) | Phase 3: Exploratory 2: PBP - CoV2 preS dTM (B.1.351) | Phase 3: Exploratory 3: PBP - CoV2 preS dTM (B.1.351) | Phase 3: Exploratory 4: PBP - CoV2 preS dTM (B.1.351)
All-Cause Mortality (participants affected / at risk) | 0/240 | 0/240 | 0/241 | 0/328 | 0/378 | 0/375 | 0/113 | 0/111 | 0/108 | 0/127 | 0/100 | 0/100 | 0/103 | 0/38 | 0/38 | 0/132 | 0/78 | 1/473 | 0/4 | 0/8 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 2/240 | 6/240 | 4/241 | 8/328 | 9/378 | 11/375 | 3/113 | 1/111 | 4/108 | 3/127 | 4/100 | 0/100 | 1/103 | 2/38 | 3/38 | 3/132 | 3/78 | 14/473 | 2/4 | 0/8 | 1/9 | 1/9
Other Adverse Events (participants affected / at risk) | 217/240 | 215/240 | 219/241 | 281/328 | 328/378 | 331/375 | 97/113 | 88/111 | 83/108 | 115/127 | 92/100 | 97/100 | 89/103 | 21/38 | 24/38 | 112/132 | 59/78 | 421/473 | 4/4 | 7/8 | 8/9 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 (N=240) | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 (N=240) | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3 (N=241) | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) (N=328) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) (N=378) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) (N=375) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) (N=113) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) (N=111) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) (N=108) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) (N=127) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) (N=100) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) (N=100) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614) (N=103) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) (N=38) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) (N=38) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) (N=132) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351) (N=78) | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614) (N=473) | Phase 3: Exploratory 1: PBP - CoV2 preS dTM (B.1.351) (N=4) | Phase 3: Exploratory 2: PBP - CoV2 preS dTM (B.1.351) (N=8) | Phase 3: Exploratory 3: PBP - CoV2 preS dTM (B.1.351) (N=9) | Phase 3: Exploratory 4: PBP - CoV2 preS dTM (B.1.351) (N=9)
Animal Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple Fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple Injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma Site Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcoholic Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervicobrachial Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss Of Consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Motor Neurone Disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trigeminal Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blindness Unilateral (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Necrotising Fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurological Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periumbilical Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pilonidal Disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis Acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum Sickness-Like Reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss Of Personal Independence In Daily Activities (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Antidepressant Discontinuation Syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis Chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus Urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 1 (N=240) | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 2 (N=240) | Phase 2: CoV2 preS dTM-AS03 (D614) Formulation 3 (N=241) | Phase 3: Cohort 1: PBP - CoV2 preS dTM-AS03 (D614) (N=328) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (B.1.351) (N=378) | Phase 3: Cohort 2: PBP - CoV2 preS dTM-AS03 (D614 + B.1.351) (N=375) | Phase 3: Cohort 1: MP - CoV2 preS dTM-AS03 (D614) (N=113) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (B.1.351) (N=111) | Phase 3: Cohort 2: MP - CoV2 preS dTM-AS03 (D614 + B.1.351) (N=108) | Phase 3: Cohort 1: OUAP - CoV2 preS dTM-AS03 (D614) (N=127) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (B.1.351) (N=100) | Phase 3: Cohort 2: OUAP - CoV2 preS dTM-AS03 (D614 + B.1.351) (N=100) | Phase 3: Cohort 1: JJJP - CoV2 preS dTM-AS03 (D614) (N=103) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (B.1.351) (N=38) | Phase 3: Cohort 2: JJJP - CoV2 preS dTM-AS03 (D614 + B.1.351) (N=38) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (D614) (N=132) | Phase 3: Cohort 2: PP - CoV2 preS dTM-AS03 (B.1.351) (N=78) | Phase 3: Comparator: CoV2 preS dTM-AS03 (D614) (N=473) | Phase 3: Exploratory 1: PBP - CoV2 preS dTM (B.1.351) (N=4) | Phase 3: Exploratory 2: PBP - CoV2 preS dTM (B.1.351) (N=8) | Phase 3: Exploratory 3: PBP - CoV2 preS dTM (B.1.351) (N=9) | Phase 3: Exploratory 4: PBP - CoV2 preS dTM (B.1.351) (N=9)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 3 (3) | 2 (2) | 5 (5) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 141 (195) | 134 (187) | 134 (198) | 130 (133) | 167 (176) | 165 (179) | 47 (49) | 50 (51) | 39 (39) | 45 (46) | 48 (51) | 55 (56) | 37 (37) | 10 (10) | 10 (10) | 51 (52) | 20 (20) | 278 (406) | 2 (2) | 3 (3) | 6 (6) | 3 (3)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (11) | 7 (8) | 8 (9) | 2 (2) | 9 (9) | 8 (8) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 26 (30) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth Impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 107 (132) | 102 (134) | 104 (131) | 91 (94) | 110 (113) | 114 (115) | 31 (32) | 39 (40) | 31 (31) | 22 (22) | 30 (30) | 35 (36) | 24 (24) | 6 (6) | 7 (7) | 42 (42) | 18 (18) | 228 (308) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 143 (196) | 135 (176) | 123 (166) | 123 (124) | 145 (148) | 153 (153) | 41 (41) | 48 (51) | 43 (43) | 40 (41) | 36 (38) | 54 (54) | 33 (33) | 9 (9) | 11 (11) | 61 (61) | 27 (27) | 275 (371) | 2 (2) | 2 (2) | 4 (4) | 4 (4)
Breast Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 5 (5) | 3 (3) | 7 (7) | 16 (16) | 34 (35) | 37 (38) | 6 (6) | 4 (4) | 9 (9) | 2 (2) | 9 (9) | 6 (6) | 5 (5) | 0 (0) | 1 (1) | 20 (20) | 13 (13) | 21 (21) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 7 (9) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis Externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 2 (2) | 7 (7) | 4 (4) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 7 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-Acute Covid-19 Syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 7 (8) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Suspected Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 3 (4) | 5 (5) | 2 (2) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 4 (4) | 3 (3) | 2 (2) | 2 (2) | 6 (6) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dust Allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 97 (113) | 93 (103) | 77 (90) | 50 (50) | 74 (75) | 77 (77) | 16 (16) | 23 (23) | 23 (23) | 23 (23) | 23 (23) | 31 (31) | 10 (10) | 5 (5) | 5 (5) | 38 (38) | 15 (15) | 160 (193) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 22 (25) | 9 (11) | 17 (19) | 9 (9) | 17 (18) | 13 (13) | 2 (2) | 3 (3) | 3 (3) | 4 (4) | 1 (1) | 6 (6) | 4 (4) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 40 (46) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection Site Erythema (General disorders) | 28 (31) | 41 (46) | 26 (29) | 32 (32) | 23 (23) | 19 (19) | 8 (8) | 7 (7) | 4 (4) | 22 (22) | 8 (8) | 9 (9) | 5 (5) | 1 (1) | 3 (3) | 9 (9) | 2 (2) | 77 (92) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection Site Pain (General disorders) | 199 (336) | 194 (331) | 200 (339) | 259 (260) | 297 (298) | 301 (302) | 89 (89) | 81 (81) | 75 (75) | 100 (100) | 86 (86) | 85 (85) | 80 (80) | 18 (18) | 19 (19) | 96 (96) | 46 (46) | 372 (590) | 4 (4) | 5 (5) | 7 (7) | 3 (3)
Injection Site Swelling (General disorders) | 40 (42) | 39 (46) | 37 (41) | 32 (33) | 37 (37) | 25 (25) | 10 (10) | 7 (7) | 4 (4) | 24 (24) | 8 (8) | 5 (5) | 6 (6) | 0 (0) | 3 (3) | 11 (11) | 3 (3) | 72 (86) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 138 (189) | 142 (183) | 146 (190) | 101 (101) | 122 (124) | 122 (126) | 42 (43) | 39 (39) | 33 (33) | 40 (40) | 35 (38) | 43 (43) | 31 (31) | 8 (8) | 7 (7) | 61 (61) | 25 (25) | 241 (331) | 1 (1) | 3 (4) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 34 (35) | 35 (36) | 29 (29) | 15 (16) | 12 (12) | 18 (19) | 1 (1) | 5 (5) | 6 (6) | 3 (3) | 4 (4) | 7 (7) | 2 (2) | 0 (0) | 1 (1) | 11 (11) | 3 (3) | 42 (44) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4) | 2 (2) | 8 (8) | 13 (14) | 12 (12) | 4 (4) | 3 (3) | 4 (4) | 7 (7) | 4 (4) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 1 (1) | 33 (36) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 4 (4) | 4 (4) | 6 (6) | 5 (5) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 13 (14) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 1 (1) | 6 (6) | 9 (10) | 11 (11) | 4 (4) | 3 (3) | 3 (3) | 2 (2) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 22 (24) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary Colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection Site Pruritus (General disorders) | 7 (7) | 14 (15) | 6 (8) | 4 (4) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 13 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT04762680/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT04762680/SAP_001.pdf